CLINICAL TRIAL: NCT00141518
Title: A Long-term Health Economics Study of Intraduodenal Levodopa (Duodopa®) in Routine Care for Patients With Advanced Idiopathic Parkinson's Disease With Severe Motor Fluctuations and Hyper-/Dyskinesia
Brief Title: Long-term Study of Duodopa (Levodopa/Carbidopa) in Advanced Parkinson's: Health Outcomes & Net Economic Impact
Acronym: DAPHNE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S187.4.001; 2005-002654-21 (EudraCT Number)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Advanced Idiopathic Parkinson's Disease
Keywords: Health economics,Quality of life
MeSH Terms: interventions — carbidopa, levodopa drug combination; Carbidopa; Jejunostomy

ARMS (3):
- Duodopa Naïve (Experimental): Duodopa-naïve participants titrated to receive Duodopa (levodopa/carbidopa intestinal gel) adjusted to an optimal clinical response for each participant, using the portable CADD Legacy Duodopa pump (CE 0473). Treatment is composed of 3 individually adjusted doses: the morning bolus dose (usually 5-10 mL [100-200 mg levodopa]); the continuous maintenance dose (usually 2-6 mL/hour [40-120 mg levodopa/hour]); and extra bolus doses, adjusted individually.
  Interventions: Drug: Levodopa-carbidopa intestinal gel (LCIG); Device: CADD-Legacy® 1400 ambulatory infusion pump; Device: percutaneous endoscopic gastrostomy tube (PEG tube); Device: jejunal extension tube (J-tube)
- Duodopa Non-naïve < 2 Years (Experimental): Duodopa non-naïve participants treated with Duodopa for < 2 years receive Duodopa (levodopa/carbidopa intestinal gel) adjusted to an optimal clinical response for each participant, using the portable CADD Legacy Duodopa pump (CE 0473). Treatment is composed of 3 individually adjusted doses: the morning bolus dose (usually 5-10 mL [100-200 mg levodopa]); the continuous maintenance dose (usually 2-6 mL/hour [40-120 mg levodopa/hour]); and extra bolus doses, adjusted individually.
  Interventions: Drug: Levodopa-carbidopa intestinal gel (LCIG); Device: CADD-Legacy® 1400 ambulatory infusion pump; Device: percutaneous endoscopic gastrostomy tube (PEG tube); Device: jejunal extension tube (J-tube)
- Duodopa Non-naïve ≥ 2 years (Experimental): Duodopa non-naïve participants treated with Duodopa for ≥ 2 years receive Duodopa (levodopa/carbidopa intestinal gel) adjusted to an optimal clinical response for each participant, using the portable CADD Legacy Duodopa pump (CE 0473). Treatment is composed of 3 individually adjusted doses: the morning bolus dose (usually 5-10 mL [100-200 mg levodopa]); the continuous maintenance dose (usually 2-6 mL/hour [40-120 mg levodopa/hour]); and extra bolus doses, adjusted individually.
  Interventions: Drug: Levodopa-carbidopa intestinal gel (LCIG); Device: CADD-Legacy® 1400 ambulatory infusion pump; Device: percutaneous endoscopic gastrostomy tube (PEG tube); Device: jejunal extension tube (J-tube)

INTERVENTIONS:
Drug: Levodopa-carbidopa intestinal gel (LCIG)
  Other Names: DUOPA™ (carbidopa and levodopa Enteral Suspension); DUODOPA®; ABT-SLV187
Device: CADD-Legacy® 1400 ambulatory infusion pump
Device: percutaneous endoscopic gastrostomy tube (PEG tube)
Device: jejunal extension tube (J-tube)

SUMMARY:
The primary objective of this study is to collect health economic data depicting the initial levels and natural progression over time of resource usage, Parkinson's disease (PD)-related costs, and health related quality of life (HRQoL) for a cohort of advanced PD patients treated with Duodopa (levodopa-carbidopa in an intestinal gel formulation), of which about one-third were Duodopa-naïve prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

- Advanced idiopathic Parkinson's disease

Exclusion Criteria:

- Other diseases which might influence compliance or participation in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-03; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bergmann, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Duodopa Naïve: Duodopa-naïve participants were titrated to receive Duodopa (levodopa/carbidopa intestinal gel) adjusted to an optimal clinical response for each participant, using the portable CADD Legacy Duodopa pump (CE 0473). Treatment is composed of 3 individually adjusted doses: the morning bolus dose (usually 5-10 mL [100-200 mg levodopa]); the continuous maintenance dose (usually 2-6 mL/hour [40-120 mg levodopa/hour]); and extra bolus doses, adjusted individually.
Period: Overall Study
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Started | 37 | 22 | 18
Safety Sample | 36 | 22 | 18
Full Analysis Sample | 27 | 22 | 18
Completed | 21 | 16 | 12
Not Completed | 16 | 6 | 6
Not completed — Withdrew Consent Prior to Treatment | 1 | 0 | 0
Not completed — Adverse Event | 7 | 5 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Lack of Efficacy | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years | Total
Number analyzed (Participants) | 27 | 22 | 18 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (6.4) | 65.4 (5.2) | 66.6 (8.7) | 65.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 6 | 24
  Male | 16 | 15 | 12 | 43

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Total Score, and UPDRS Subscores I, II, III, and IV at Baseline and Month 12
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. For Parts I-III and Total Score, each question is measured on a 5-point scale of 0 (normal or no disease effect) to 4 (maximum negative effect); for Part IV, questions are measured on a 5- or 2-point scale (0 or 1). Part I score is the sum of answers to 'Mentation, Behavior and Mood' questions, with a score range from 0-16. Part II score is the sum of answers to 'Activities of Daily Living' questions, with a score range from 0-52. Part III score is the sum of answers to 'Motor Examination' questions, with a score range from 0-108. Part IV score is the sum of answers to 'Complications of Therapy' questions, with a score range from 0-23. Total Score is the sum of the responses to the 31 questions (44 answers) that comprise Parts I-III of the scale, with a score range from 0-176. Higher scores are associated with more disability.
Time Frame: Baseline (Month -3), Month 12
Population: Full Analysis Set: Participants who had ≥1 dose of study drug and (for Duodopa naives) data for baseline (BL) and ≥1 post-BL assessment of the primary efficacy measurements UPDRS and EQ-5D or (for Duodopa non-naives) had data for Month 0 visit and ≥1 more assessment of UPDRS and EQ-5D. n=participants with assessments at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Total Score, Baseline (Month -3); n=27, 0, 0 | 52.1 (16.1) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Total Score, Month 12; n=25, 20, 17 | 42.5 (22.6) | 44.0 (13.9) | 48.2 (18.4)
  Part I, Baseline (Month -3); n=27, 0, 0 | 2.9 (1.9) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Part I, Month 12; n=25, 20, 17 | 3.1 (2.2) | 2.6 (2.0) | 3.2 (2.2)
  Part II, Baseline (Month -3); n=27, 0, 0 | 15.4 (5.7) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Part II, Month 12; n=25, 20, 17 | 12.2 (6.8) | 13.4 (5.7) | 14.3 (6.0)
  Part III, Baseline (Month -3); n=27, 0, 0 | 24.4 (11.0) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Part III, Month 12; n=25, 20, 17 | 21.5 (13.2) | 21.2 (10.0) | 23.5 (11.5)
  Part IV, Baseline (Month -3); n=27, 0, 0 | 9.4 (2.6) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Part IV, Month 12; n=25, 20, 17 | 5.7 (3.4) | 7.0 (2.5) | 7.2 (3.5)
Statistical Analysis 1: Comparison: Duodopa Naïve; Total Score, Change From Baseline for the Duodopa Naïve group at Month 12 (n=25); Test type: Superiority or Other; p = 0.017, Wilcoxon tests; mean change from baseline = -9.4, Standard Deviation 17.5

2. Primary Outcome: Euro QoL 5 Dimensions Quality of Life Instrument (EQ-5D) Descriptive Systems Summary Index Score at Baseline and Month 12
Description: The EQ-5D is a participant-answered questionnaire scoring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that essentially attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.11 (worst health state) to 1.00 (perfect health state).
Time Frame: Baseline (Month -3), Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 0.57 (0.26) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 12; n=25, 20, 17 | 0.59 (0.33) | 0.66 (0.36) | 0.51 (0.37)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 12 (n=25); Test type: Superiority or Other; p = 0.919, Wilcoxon tests; mean change from baseline = 0.02, Standard Deviation 0.29

3. Primary Outcome: EQ-5D Visual Analog Scale (VAS) Score at Baseline and Month 12
Description: The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where 100 is the 'best imaginable health state' and 0 is the 'worst imaginable health state.' The scale was normalized to a scale of 0 to 1, with higher values indicating a better health state.
Time Frame: Baseline (Month -3), Month 12
Population: Full Analysis Set: Participants who had ≥ 1 dose of study medication and (for Duodopa naives) had data for baseline and ≥ 1 post-baseline assessment of the primary efficacy measurements UPDRS and EQ-5D or (for Duodopa non-naives) had data for Month 0 visit and ≥ 1 more assessment of the primary efficacy measurements UPDRS and EQ-5D.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 0.44 (0.20) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 12; n=25, 19, 17 | 0.63 (0.18) | 0.64 (0.19) | 0.64 (0.22)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 12 (n=25); Test type: Superiority or Other; p = 0.002, Wilcoxon tests; mean change from baseline = 0.18, Standard Deviation 0.24

4. Primary Outcome: Total Monthly Cost Per Participant, in Swedish Crowns (SEK) 2010
Description: Total monthly costs include
  * Direct medical costs (inpatient care, outpatient care, and drug costs [including Duodopa cost and cost of concomitant anti-PD medication]).
  * Direct non-medical costs (nursing home, home help, personal assistance, informal care [from family member or friend] and transportation to inpatient, outpatient visits and nursing home).
  * Indirect costs (sick-leave and early retirement due to PD [applied to individuals only up to the age of 65 since the main indirect cost item, early retirement due to disability, is only available for individuals 30-64 years old. Sixty-five is also a common retirement age in Sweden]).
  The average rate for US Dollar (USD) to SEK on 31 December 2010 was 1 USD = 6.734 SEK.
Time Frame: Baseline (month -3) for Duodopa-naïve participants, then at Month 0, and monthly thereafter until study completion (up to 48 months) for all participants
Measure: Mean (Standard Deviation); unit: SEK 2010
Units Other Than Participants: Patient-months per Study Arm
Groups:
- Total: All participants
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years | Total
Number analyzed (Participants) | 37 | 22 | 18 | 77
Number analyzed (Patient-months per Study Arm) | 920 | 710 | 574 | 2204
SEK 2010 | 78418 (42028) | 75521 (73296) | 82177 (53728) | 78464 (56772)

5. Primary Outcome: Monthly Drug Costs Per Participant, SEK 2010
Description: Drug costs include Duodopa cost and cost of concomitant anti-PD medication. Drug costs are a direct medical cost. The average rate for US Dollar (USD) to SEK on 31 December 2010 was 1 USD = 6.734 SEK.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: SEK 2010
Units Other Than Participants: Patient-months per Study Arm
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years | Total
Number analyzed (Participants) | 37 | 22 | 18 | 77
Number analyzed (Patient-months per Study Arm) | 920 | 710 | 574 | 2204
SEK 2010 | 39382 (16733) | 34417 (10494) | 37679 (15196) | 37339 (14725)

6. Primary Outcome: Monthly Direct Medical Cost (Excluding Drug Costs) Per Participant, SEK 2010
Description: Direct medical costs consist of inpatient care, outpatient care (visits to physician, nurse, physiotherapist, occupational therapist, dietitian, speech therapist, counselor, and phone consultations). The average rate for US Dollar (USD) to SEK on 31 December 2010 was 1 USD = 6.734 SEK.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: SEK 2010
Units Other Than Participants: Patient-months per Study Arm
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years | Total
Number analyzed (Participants) | 37 | 22 | 18 | 77
Number analyzed (Patient-months per Study Arm) | 920 | 710 | 574 | 2204
SEK 2010 | 3825 (9394) | 4552 (11819) | 3607 (8648) | 4002 (10069)

7. Primary Outcome: Direct Monthly Non-medical Costs Per Participant, SEK 2010
Description: Direct non-medical costs include nursing home, home help, personal assistance, informal care (from family member or friend) and transportation to inpatient, outpatient visits and nursing home. The average rate for US Dollar (USD) to SEK on 31 December 2010 was 1 USD = 6.734 SEK.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: SEK 2010
Units Other Than Participants: Patient-months per Study Arm
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years | Total
Number analyzed (Participants) | 37 | 22 | 18 | 77
Number analyzed (Patient-months per Study Arm) | 920 | 710 | 574 | 2204
SEK 2010 | 19274 (26485) | 27439 (61656) | 25008 (42455) | 23398 (44698)

8. Primary Outcome: Indirect Monthly Costs Per Participant (Only Applied to Participants Younger Than 65) by Study Month, SEK 2010
Description: Indirect costs consist of sick-leave and early retirement due to PD, are applied to individuals only up to the age of 65 since the main indirect cost item - early retirement due to disability - is only available for individuals 30-64 years old. Sixty-five is also a common retirement age in Sweden. The average rate for US Dollar (USD) to SEK on 31 December 2010 was 1 USD = 6.734 SEK.
Time Frame: Baseline (month -3) for Duodopa-naïve participants, then at Month 0, and monthly thereafter until Month 36
Population: All participants; n=fraction of number of participants younger than 65 years with indirect costs / number of participants assessed at given time point.
Measure: Mean (Standard Deviation); unit: SEK 2010
Groups:
- Total: Duodopa-naïve participants, Duodopa non-naïve participants treated with Duodopa for < 2 years, and Duodopa non-naïve participants treated with Duodopa for ≥ 2 years received Duodopa (levodopa/carbidopa intestinal gel) adjusted to an optimal clinical response for each participant, using the portable CADD Legacy Duodopa pump (CE 0473). Treatment is composed of 3 individually adjusted doses: the morning bolus dose (usually 5-10 mL [100-200 mg levodopa]); the continuous maintenance dose (usually 2-6 mL/hour [40-120 mg levodopa/hour]); and extra bolus doses, adjusted individually.
Arm/Group | Total
Number analyzed (Participants) | 77
SEK 2010
  Month -3; n=15/37 | 17032 (20911)
  Month 0; n=23/67 | 14109 (19823)
  Month 1; n=23/67 | 14109 (19823)
  Month 2; n=22/65 | 13896 (19746)
  Month 3; n=23/65 | 14543 (19971)
  Month 4; n=23/65 | 14543 (19971)
  Month 5; n=22/65 | 13896 (19746)
  Month 6; n=21/65 | 13250 (19498)
  Month 7; n=24/65 | 15512 (20433)
  Month 8; n=24/63 | 16005 (20566)
  Month 9; n=22/62 | 14569 (19978)
  Month 10; n=22/62 | 14569 (19978)
  Month 11; n=22/62 | 14399 (19785)
  Month 12; n=22/62 | 14399 (19785)
  Month 13; n=22/62 | 14230 (19681)
  Month 14; n=22/62 | 14569 (19978)
  Month 15; n=22/61 | 14808 (20055)
  Month 16; n=22/61 | 14808 (20055)
  Month 17; n=22/61 | 14463 (19758)
  Month 18; n=22/61 | 14463 (19758)
  Month 19; n=22/60 | 14704 (19834)
  Month 20; n=20/59 | 13529 (19411)
  Month 21; n=20/58 | 13763 (19497)
  Month 22; n=18/57 | 12530 (18980)
  Month 23; n=18/57 | 12530 (18980)
  Month 24; n=17/56 | 12003 (18727)
  Month 25; n=16/54 | 12059 (18966)
  Month 26; n=18/54 | 13615 (19637)
  Month 27; n=16/53 | 12683 (19471)
  Month 28; n=15/53 | 11890 (19106)
  Month 29; n=16/53 | 12683 (19471)
  Month 30; n=16/53 | 12683 (19471)
  Month 31; n=15/50 | 12604 (19448)
  Month 32; n=14/50 | 11763 (19055)
  Month 33; n=14/50 | 11763 (19055)
  Month 34; n=14/49 | 12003 (19176)
  Month 35; n=14/49 | 12003 (19176)
  Month 36; n=15/49 | 12432 (19137)

9. Secondary Outcome: Modified Hoehn and Yahr Staging: Current Stage From Baseline to Month 36
Description: The current stage of PD was characterized according to Modified Hoehn and Yahr criteria, measured on the following 8-point scale for staging: 0=no signs of disease; 1=unilateral disease; 1.5=unilateral plus axial involvement; 2=bilateral disease; 2.5=mild bilateral disease; 3=mild to moderate bilateral disease; 4=severe disability; and 5=wheelchair bound or bedridden unless aided.
Time Frame: Baseline (Month -3), Months 0, 3, 6, 9, 12, 18, 24, 30, 36, endpoint (last non-missing value assigned to treatment for the participant)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 2.7 (0.7) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 2.5 (0.7) | 2.7 (0.8) | 3.2 (0.8)
  Month 3; n=24, 22, 18 | 2.3 (0.8) | 2.7 (0.8) | 3.0 (0.8)
  Month 6; n=25, 22, 18 | 2.4 (0.8) | 2.6 (0.9) | 3.1 (0.8)
  Month 9; n=25, 20, 17 | 2.4 (1.0) | 2.7 (0.7) | 3.1 (0.7)
  Month 12; n=25, 20, 17 | 2.4 (0.8) | 2.8 (0.7) | 3.3 (0.8)
  Month 18; n=24, 20, 17 | 2.4 (0.9) | 2.7 (0.7) | 3.4 (1.0)
  Month 24; 23, 18, 15 | 2.5 (0.9) | 3.0 (0.9) | 3.2 (0.8)
  Month 30; n=23, 17, 13 | 2.7 (1.1) | 2.9 (0.8) | 3.1 (0.9)
  Month 36; n=21, 16, 12 | 2.7 (1.2) | 2.9 (0.6) | 3.3 (0.9)
  Endpoint; n=27, 22, 18 | 2.7 (1.1) | 3.1 (0.8) | 3.4 (0.8)

10. Secondary Outcome: Modified Hoehn and Yahr Staging: Best Stage From Baseline to Month 36
Description: The best PD stage that the participant experienced during the last month was characterized according to Modified Hoehn and Yahr criteria, measured on the following 8-point scale for staging: 0=no signs of disease; 1=unilateral disease; 1.5=unilateral plus axial involvement; 2=bilateral disease; 2.5=mild bilateral disease; 3=mild to moderate bilateral disease; 4=severe disability; and 5=wheelchair bound or bedridden unless aided.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 2.2 (1.2) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 2.0 (0.9) | 2.5 (0.7) | 2.5 (0.7)
  Month 3; n=24, 22, 18 | 2.0 (0.9) | 2.5 (0.6) | 2.6 (0.8)
  Month 6; n=25, 22, 18 | 2.0 (0.8) | 2.5 (0.7) | 2.6 (0.9)
  Month 9; 25, 20, 17 | 2.2 (1.1) | 2.5 (0.7) | 2.7 (0.7)
  Month 12; n=25, 20, 17 | 2.2 (0.8) | 2.6 (0.9) | 2.9 (0.8)
  Month 18; n=24, 20, 17 | 2.2 (0.9) | 2.5 (0.9) | 2.9 (0.9)
  Month 24; n=23, 18, 15 | 2.3 (1.1) | 2.6 (1.0) | 2.9 (0.8)
  Month 30; n=23, 17, 13 | 2.5 (1.2) | 2.6 (1.0) | 3.0 (0.9)
  Month 36; n=21, 16, 12 | 2.5 (1.3) | 2.6 (0.6) | 3.0 (0.7)
  Endpoint; n=27, 22, 18 | 2.6 (1.2) | 2.7 (0.7) | 3.1 (0.8)

11. Secondary Outcome: Modified Hoehn and Yahr Staging: Worst Stage From Baseline to Month 36
Description: The worst PD stage that the participant experienced during the last month was characterized according to Modified Hoehn and Yahr criteria, measured on the following 8-point scale for staging: 0=no signs of disease; 1=unilateral disease; 1.5=unilateral plus axial involvement; 2=bilateral disease; 2.5=mild bilateral disease; 3=mild to moderate bilateral disease; 4=severe disability; and 5=wheelchair bound or bedridden unless aided.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 3.8 (1.0) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 3.6 (1.1) | 3.7 (0.9) | 4.0 (0.6)
  Month 3; n=24, 22, 18 | 3.8 (1.2) | 3.7 (0.9) | 4.1 (0.7)
  Month 6; n=25, 22, 18 | 3.7 (1.3) | 3.7 (1.1) | 4.0 (0.7)
  Month 9; n=25, 20, 17 | 3.7 (1.2) | 3.8 (0.7) | 4.0 (0.5)
  Month 12; n=25, 20, 17 | 3.6 (1.3) | 3.8 (0.8) | 4.2 (0.5)
  Month 18; n=24, 20, 17 | 3.8 (1.3) | 3.9 (0.8) | 4.3 (0.6)
  Month 24; n=23, 18, 15 | 3.9 (1.3) | 3.8 (0.8) | 4.4 (0.5)
  Month 30; n=23, 17, 13 | 4.0 (1.1) | 4.0 (0.8) | 4.5 (0.7)
  Month 36; n=21, 16, 12 | 3.9 (1.2) | 4.0 (0.6) | 4.6 (0.5)
  Endpoint; n=27, 22, 18 | 3.9 (1.1) | 4.0 (0.7) | 4.5 (0.5)

12. Secondary Outcome: Schwab and England Scale: Best "On" Period Stage From Baseline to Month 36
Description: The Schwab and England scale was used to rate the subject's best "on" period during the past week by recording the percentage score, ranging between being completely independent (100%) and totally dependent (10%). "On" time is when PD symptoms are well controlled by the drug.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage score on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
percentage score on a scale
  Baseline (Month -3); n=27, 0, 0 | 74.4 (15.8) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 80.4 (13.2) | 75.5 (14.4) | 74.4 (11.5)
  Month 3; n=24, 22, 18 | 77.9 (14.4) | 75.9 (14.4) | 72.2 (15.2)
  Month 6; n=25, 22, 18 | 75.2 (15.3) | 77.3 (11.6) | 72.2 (12.6)
  Month 9; n=25, 20, 17 | 79.2 (13.5) | 76.5 (13.1) | 70.6 (13.0)
  Month 12; n=25, 20, 17 | 77.2 (13.4) | 72.5 (15.9) | 71.8 (12.4)
  Month 18; n=24, 20, 17 | 75.8 (12.8) | 74.0 (11.9) | 69.4 (14.3)
  Month 24; n=23, 18, 15 | 72.2 (18.1) | 73.3 (14.6) | 68.0 (15.2)
  Month 30; n=23, 17, 13 | 70.4 (18.7) | 71.8 (16.7) | 67.7 (17.9)
  Month 36; n=21, 16, 12 | 66.7 (21.1) | 73.1 (13.0) | 64.2 (21.1)
  Endpoint; n=27, 22, 18 | 68.9 (19.5) | 71.4 (13.2) | 62.2 (17.7)

13. Secondary Outcome: Mini Mental Status Examination (MMSE) Total Scores From Baseline to Month 36
Description: The MMSE is used to assess orientation, attention, immediate and short term recall, language, and ability to follow simple verbal and written commands. The test consists of five sections (orientation, registration, attention-calculation, recall, and language) and results in a total possible score of 0 to 30, with higher scores indicating better function.
Time Frame: Baseline (Month -3), Months 0, 3, 6, 9, 12, 18, 24, 30, 36, endpoint visit (Month 36 or last visit if discontinued early)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 28.2 (2.2) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 27.8 (2.4) | 28.0 (2.2) | 28.2 (1.4)
  Month 3; n=24, 22, 18 | 28.0 (2.9) | 27.2 (2.8) | 28.6 (1.9)
  Month 6; n=25, 21, 18 | 28.1 (2.5) | 27.6 (1.9) | 28.1 (1.4)
  Month 9; n=25, 20, 17 | 28.4 (2.3) | 27.6 (2.0) | 28.3 (2.1)
  Month 12; n=25, 20, 17 | 27.9 (2.8) | 28.2 (1.7) | 28.2 (2.5)
  Month 18; n=24, 19, 16 | 27.6 (2.7) | 28.5 (1.4) | 28.3 (2.3)
  Month 24; n=23, 18, 15 | 27.7 (2.5) | 27.8 (2.0) | 28.0 (2.2)
  Month 30; n=23, 17, 13 | 27.3 (3.9) | 26.4 (3.4) | 28.6 (2.0)
  Month 36; n=21, 16, 12 | 27.2 (3.2) | 26.3 (4.0) | 27.9 (4.1)
  Endpoint; n=27, 22, 17 | 27.1 (3.9) | 26.4 (3.8) | 27.3 (3.8)

14. Secondary Outcome: MMSE Orientation Subscale Scores From Baseline to Month 36
Description: The MMSE is used to assess orientation, attention, immediate and short term recall, language, and ability to follow simple verbal and written commands. The orientation subscale has a total possible score of 0 to 10, with higher scores indicating better function.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 9.8 (0.6) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 9.6 (1.1) | 9.9 (0.4) | 9.8 (0.4)
  Month 3; n=24, 22, 18 | 9.4 (1.2) | 9.5 (1.1) | 9.6 (0.6)
  Month 6; n=25, 21, 18 | 9.7 (0.7) | 9.6 (0.9) | 9.7 (0.6)
  Month 9; n=25, 20, 17 | 9.8 (0.5) | 9.9 (0.4) | 9.6 (1.0)
  Month 12; n=25, 20, 17 | 9.6 (1.1) | 9.8 (0.6) | 9.7 (1.0)
  Month 18; n=24, 19, 16 | 9.7 (0.7) | 9.7 (0.6) | 9.9 (0.3)
  Month 24; n=23, 18, 15 | 9.7 (0.6) | 9.8 (0.5) | 9.9 (0.4)
  Month 30; n=23, 17, 13 | 9.4 (1.2) | 8.9 (1.9) | 9.8 (0.6)
  Month 36; n=21, 16, 12 | 9.6 (1.0) | 9.3 (1.2) | 9.1 (2.2)
  Endpoint; n=27, 22, 17 | 9.5 (1.1) | 8.9 (1.6) | 9.2 (1.8)

15. Secondary Outcome: MMSE Registration Subscale Scores From Baseline to Month 36
Description: The MMSE is used to assess orientation, attention, immediate and short term recall, language, and ability to follow simple verbal and written commands. The Registration subscale a total possible score of 0 to 3, with higher scores indicating better function.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 3.0 (0.0) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 3.0 (0.2) | 3.0 (0.2) | 3.0 (0.0)
  Month 3; n=24, 22, 18 | 3.0 (0.0) | 3.0 (0.2) | 3.0 (0.0)
  Month 6; n=25, 21, 18 | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0)
  Month 9; n=25, 20, 17 | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0)
  Month 12; n=25, 20, 17 | 3.0 (0.2) | 3.0 (0.0) | 3.0 (0.0)
  Month 18; n=24, 19, 16 | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0)
  Month 24; n=23, 18, 15 | 3.0 (0.2) | 3.0 (0.0) | 3.0 (0.0)
  Month 30; n=23, 17, 13 | 3.0 (0.0) | 2.9 (0.2) | 3.0 (0.0)
  Month 36; n=21, 16, 12 | 3.0 (0.0) | 3.0 (0.0) | 2.9 (0.3)
  Endpoint; n=27, 22, 17 | 3.0 (0.0) | 3.0 (0.0) | 2.9 (0.2)

16. Secondary Outcome: MMSE Attention and Calculation Subscale Scores From Baseline to Month 36
Description: The MMSE is used to assess orientation, attention, immediate and short term recall, language, and ability to follow simple verbal and written commands. The Attention and Calculation subscale results in a total possible score of 0 to 5, with higher scores indicating better function.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 4.9 (0.4) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 4.6 (0.9) | 4.4 (1.4) | 4.6 (0.7)
  Month 3; n=24, 22, 18 | 4.6 (0.9) | 4.3 (1.3) | 4.7 (0.8)
  Month 6; n=25, 21, 18 | 4.6 (1.0) | 4.5 (0.8) | 4.7 (0.6)
  Month 9; n=25, 20, 17 | 4.7 (0.6) | 4.3 (1.0) | 4.8 (0.5)
  Month 12; n=25, 20, 17 | 4.7 (0.6) | 4.7 (0.7) | 4.6 (0.7)
  Month 18; n=24, 19, 16 | 4.5 (1.1) | 4.7 (0.8) | 4.5 (1.1)
  Month 24; n=23, 18, 15 | 4.6 (0.7) | 4.6 (0.6) | 4.3 (1.2)
  Month 30; n=23, 17, 13 | 4.6 (1.0) | 4.1 (1.2) | 4.8 (0.4)
  Month 36; n=21, 16, 12 | 4.2 (1.5) | 3.7 (1.9) | 4.8 (0.6)
  Endpoint; n=27, 22, 17 | 4.2 (1.5) | 4.0 (1.7) | 4.4 (0.9)

17. Secondary Outcome: MMSE Recall Subscale Scores From Baseline to Month 36
Description: The MMSE is used to assess orientation, attention, immediate and short term recall, language, and ability to follow simple verbal and written commands. The Recall subscale results in a total possible score of 0 to 3, with higher scores indicating better function.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 2.2 (0.9) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 2.2 (1.0) | 2.1 (0.8) | 2.3 (0.8)
  Month 3; n=24, 22, 18 | 2.5 (0.9) | 2.1 (0.9) | 2.5 (0.6)
  Month 6; n=25, 21, 18 | 2.5 (0.8) | 2.4 (0.8) | 2.3 (0.8)
  Month 9; n=25, 20, 17 | 2.5 (0.8) | 2.2 (0.8) | 2.5 (0.9)
  Month 12; n=25, 20, 17 | 2.5 (0.9) | 2.5 (0.8) | 2.6 (0.9)
  Month 18; n=24, 19, 16 | 2.3 (0.7) | 2.5 (0.5) | 2.6 (0.9)
  Month 24; n=23, 18, 15 | 2.4 (0.8) | 2.3 (0.8) | 2.5 (0.9)
  Month 30; n=23, 17, 13 | 2.5 (0.9) | 2.5 (0.6) | 2.6 (0.8)
  Month 36; n=21, 16, 12 | 2.2 (0.9) | 2.4 (0.7) | 2.8 (0.5)
  Endpoint; n=27, 22, 17 | 2.2 (0.9) | 2.5 (0.7) | 2.5 (0.8)

18. Secondary Outcome: MMSE Language Subscale Scores From Baseline to Month 36
Description: The MMSE is used to assess orientation, attention, immediate and short term recall, language, and ability to follow simple verbal and written commands. The Language subscale results in a total possible score of 0 to 9, with higher scores indicating better function.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 8.3 (1.6) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 8.5 (0.9) | 8.6 (0.5) | 8.5 (0.7)
  Month 3; n=24, 22, 18 | 8.4 (0.7) | 8.3 (0.9) | 8.7 (0.5)
  Month 6; n=25, 21, 18 | 8.3 (0.9) | 8.1 (1.3) | 8.3 (0.7)
  Month 9; n=25, 20, 17 | 8.4 (1.0) | 8.2 (0.9) | 8.4 (0.7)
  Month 12; n=25, 20, 17 | 8.2 (1.3) | 8.3 (0.7) | 8.2 (0.8)
  Month 18; n=24, 19, 16 | 8.2 (1.1) | 8.6 (0.6) | 8.3 (0.9)
  Month 24; n=23, 18, 15 | 8.0 (1.4) | 8.1 (0.9) | 8.3 (0.8)
  Month 30; n=23, 17, 13 | 7.9 (1.4) | 8.0 (0.9) | 8.5 (1.0)
  Month 36; n=21, 16, 12 | 8.3 (0.9) | 7.9 (1.3) | 8.4 (1.0)
  Endpoint; n=27, 22, 17 | 8.3 (0.9) | 7.9 (1.3) | 8.4 (1.0)

19. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS) Total Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Total score ranges from 0 (no depression) to 60 (severely depressed).
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 28
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 10.3 (5.6) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 9.0 (5.3) | 7.8 (5.2) | 8.8 (5.8)
  Month 3; n=24, 22, 17 | 10.2 (6.3) | 8.1 (4.9) | 8.4 (5.8)
  Month 6; n=25, 21, 17 | 10.5 (6.9) | 8.4 (3.8) | 8.5 (5.3)
  Month 9; n=25, 20, 17 | 8.8 (4.9) | 8.0 (3.4) | 9.9 (6.5)
  Month 12; n=25, 20, 17 | 8.6 (5.7) | 8.8 (5.2) | 9.5 (7.3)
  Month 18; n=24, 19, 16 | 10.6 (6.2) | 8.1 (4.5) | 9.1 (7.1)
  Month 24; n=23, 18, 15 | 10.1 (5.6) | 9.7 (5.5) | 11.1 (7.4)
  Month 30; n=22, 17, 13 | 12.0 (5.9) | 10.6 (4.6) | 9.0 (5.0)
  Month 36; n=21, 16, 12 | 12.2 (7.3) | 9.1 (4.5) | 10.4 (9.4)
  Endpoint; n=26, 22, 17 | 11.6 (7.0) | 9.0 (4.9) | 12.3 (9.1)

20. Secondary Outcome: MADRS Reported Sadness Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Reported Sadness scores rate depressed mood, regardless of whether it is reflected in appearance or not, and includes low spirits, despondency or the feeling of being beyond help and without hope.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 0.9 (0.8) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 0.6 (0.7) | 0.8 (1.2) | 0.8 (1.0)
  Month 3; n=24, 22, 17 | 0.9 (1.0) | 0.6 (0.8) | 0.5 (0.6)
  Month 6; n=25, 21, 17 | 1.1 (1.1) | 0.8 (0.6) | 0.5 (0.7)
  Month 9; n=25, 20, 17 | 0.9 (0.7) | 0.9 (0.8) | 1.1 (1.4)
  Month 12; n=25, 20, 17 | 0.6 (0.7) | 1.1 (0.9) | 0.8 (1.0)
  Month 18; n=24, 19, 16 | 1.0 (1.0) | 0.7 (0.7) | 0.8 (0.8)
  Month 24; n=23, 18, 15 | 1.0 (1.0) | 0.9 (0.9) | 0.8 (0.7)
  Month 30; n=23, 17, 13 | 1.2 (0.9) | 0.9 (0.8) | 0.9 (1.0)
  Month 36; n=21, 16, 12 | 1.1 (1.2) | 0.9 (0.9) | 1.1 (1.1)
  Endpoint; n=27, 22, 17 | 1.2 (1.2) | 0.8 (0.9) | 1.0 (1.0)

21. Secondary Outcome: MADRS Apparent Sadness Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Apparent sadness scores rate despondency, gloom and despair (more than just ordinary transient low spirits), reflected in speech, facial expression, and posture.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 0.7 (0.8) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 0.4 (0.8) | 0.5 (0.9) | 0.8 (0.7)
  Month 3; n=24, 22, 17 | 0.8 (0.9) | 0.6 (0.8) | 0.5 (0.7)
  Month 6; n=25, 21, 17 | 1.0 (1.1) | 0.6 (0.5) | 0.5 (0.6)
  Month 9; n=25, 20, 17 | 0.9 (0.8) | 0.7 (0.7) | 0.9 (1.0)
  Month 12; n=25, 20, 17 | 0.4 (0.5) | 0.9 (1.0) | 0.8 (0.8)
  Month 18; n=24, 19, 16 | 0.8 (0.9) | 0.6 (0.7) | 0.8 (0.9)
  Month 24; n=23, 18, 15 | 1.0 (1.2) | 0.6 (0.7) | 0.7 (0.6)
  Month 30; n=23, 17, 13 | 1.2 (1.0) | 1.0 (0.9) | 0.6 (0.7)
  Month 36; n=21, 16, 12 | 1.1 (1.2) | 0.8 (0.9) | 1.3 (1.4)
  Endpoint; n=27, 22, 17 | 1.1 (1.2) | 0.8 (1.0) | 1.0 (1.2)

22. Secondary Outcome: MADRS Inner Tension Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Inner Tension scores rate feelings of ill-defined discomfort, edginess, inner turmoil, mental tension mounting to either panic, dread or anguish.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 1.3 (1.3) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 1.3 (1.1) | 1.0 (1.0) | 0.9 (1.0)
  Month 3; n=24, 22, 17 | 1.5 (1.3) | 0.8 (1.0) | 0.9 (1.0)
  Month 6; n=25, 21, 17 | 1.1 (1.1) | 0.9 (1.0) | 1.2 (1.1)
  Month 9; n=25, 20, 17 | 0.9 (1.2) | 0.6 (0.8) | 0.9 (1.1)
  Month 12; n=25, 20, 17 | 1.1 (1.1) | 0.7 (0.9) | 1.5 (1.0)
  Month 18; n=24, 19, 16 | 1.2 (1.1) | 0.7 (0.9) | 0.8 (1.0)
  Month 24; n=23, 18, 15 | 1.0 (1.1) | 0.8 (1.1) | 1.3 (1.3)
  Month 30; n=23, 17, 13 | 1.1 (1.1) | 1.1 (1.2) | 1.5 (1.1)
  Month 36; n=21, 16, 12 | 1.7 (1.2) | 0.6 (0.8) | 1.3 (1.2)
  Endpoint; n=27, 22, 17 | 1.6 (1.1) | 0.6 (0.8) | 1.5 (1.3)

23. Secondary Outcome: MADRS Reduced Sleep Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Reduced Sleep scores rate the experience of reduced duration or depth of sleep compared to the participant's own normal pattern when well.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 2.5 (1.7) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 1.9 (1.6) | 1.5 (1.6) | 1.7 (1.8)
  Month 3; n=24, 22, 17 | 2.0 (1.4) | 1.8 (1.6) | 1.2 (1.2)
  Month 6; n=25, 21, 17 | 1.8 (1.8) | 1.7 (1.5) | 1.5 (1.7)
  Month 9; n=25, 20, 17 | 1.8 (1.5) | 1.9 (1.3) | 1.4 (1.5)
  Month 12; n=25, 20, 17 | 1.8 (1.5) | 1.5 (1.5) | 1.2 (1.4)
  Month 18; n=24, 19, 16 | 1.7 (1.3) | 1.5 (1.5) | 1.7 (1.4)
  Month 24; n=23, 18, 15 | 1.6 (1.3) | 1.8 (1.9) | 1.5 (1.7)
  Month 30; n=23, 17, 13 | 2.3 (1.7) | 1.9 (1.9) | 0.9 (1.0)
  Month 36; n=21, 16, 12 | 1.9 (1.7) | 1.2 (1.4) | 1.2 (1.5)
  Endpoint; n=27, 22, 17 | 1.6 (1.7) | 1.4 (1.5) | 2.0 (2.2)

24. Secondary Outcome: MADRS Reduced Appetite Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Reduced Appetite scores rate the feeling of a loss of appetite compared with when-well. Rate by loss of desire for food or the need to force oneself to eat.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 0.8 (1.1) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 0.6 (0.8) | 0.2 (0.5) | 0.3 (0.8)
  Month 3; n=24, 22, 17 | 0.7 (1.0) | 0.4 (0.8) | 0.4 (1.0)
  Month 6; n=25, 21, 17 | 0.8 (1.1) | 0.3 (0.7) | 0.5 (1.2)
  Month 9; n=25, 20, 17 | 0.5 (0.8) | 0.4 (0.6) | 0.8 (1.4)
  Month 12; n=25, 20, 17 | 0.5 (0.8) | 0.6 (0.8) | 0.7 (1.2)
  Month 18; n=24, 19, 16 | 0.5 (0.8) | 0.3 (0.7) | 0.4 (0.9)
  Month 24; n=23, 18, 15 | 0.7 (1.2) | 0.5 (0.8) | 0.7 (1.1)
  Month 30; n=23, 17, 13 | 1.0 (1.2) | 0.4 (0.6) | 0.5 (1.1)
  Month 36; n=21, 16, 12 | 0.9 (1.2) | 0.4 (0.7) | 1.1 (1.4)
  Endpoint; n=27, 22, 17 | 0.9 (1.2) | 0.3 (0.6) | 1.1 (1.3)

25. Secondary Outcome: MADRS Concentration Difficulties Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Concentration Difficulties scores rate difficulties in collecting one's thoughts mounting to an incapacitating lack of concentration.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 1.0 (1.0) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 1.0 (1.2) | 1.5 (1.3) | 0.9 (1.2)
  Month 3; n=24, 22, 17 | 0.9 (1.1) | 1.3 (0.9) | 1.2 (1.2)
  Month 6; n=25, 21, 17 | 1.2 (1.2) | 1.4 (0.9) | 1.2 (1.1)
  Month 9; n=25, 20, 17 | 1.0 (1.2) | 1.1 (1.1) | 1.3 (1.2)
  Month 12; n=25, 20, 17 | 0.9 (1.2) | 1.2 (1.1) | 1.4 (1.3)
  Month 18; n=24, 19, 16 | 1.5 (1.4) | 1.4 (1.0) | 1.4 (1.3)
  Month 24; n=23, 18, 15 | 1.5 (1.3) | 1.7 (1.5) | 1.7 (1.4)
  Month 30; n=23, 17, 13 | 1.5 (1.7) | 2.1 (1.1) | 1.5 (1.5)
  Month 36; n=21, 16, 12 | 1.6 (1.3) | 1.9 (1.3) | 1.2 (1.7)
  Endpoint; n=27, 22, 17 | 1.6 (1.5) | 1.7 (1.3) | 1.6 (1.7)

26. Secondary Outcome: MADRS Lassitude Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Lassitude scores rate difficulty in getting started or slowness in initiating and performing everyday activities.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 1.3 (1.4) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 1.4 (1.3) | 1.4 (1.2) | 1.7 (1.5)
  Month 3; n=24, 22, 17 | 1.7 (1.3) | 1.5 (1.0) | 2.0 (1.6)
  Month 6; n=25, 21, 17 | 1.5 (1.3) | 1.5 (1.2) | 1.3 (1.5)
  Month 9; n=25, 20, 17 | 1.3 (1.2) | 1.5 (1.2) | 1.7 (1.2)
  Month 12; n=25, 20, 17 | 1.6 (1.4) | 1.6 (1.3) | 1.4 (1.6)
  Month 18; n=24, 19, 16 | 1.8 (1.6) | 1.4 (1.2) | 1.6 (1.1)
  Month 24; n=23, 18, 15 | 1.7 (1.5) | 1.9 (1.1) | 1.7 (1.4)
  Month 30; n=23, 17, 13 | 2.0 (1.4) | 1.7 (1.3) | 1.3 (1.1)
  Month 36; n=21, 16, 12 | 1.9 (1.5) | 1.8 (1.4) | 1.7 (1.4)
  Endpoint; n=27, 22, 17 | 1.8 (1.5) | 1.7 (1.4) | 1.7 (1.4)

27. Secondary Outcome: MADRS Inability to Feel Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Inability to Feel scores rate the subjective experience of reduced interest in the surroundings, or activities that normally give pleasure. The ability to react with adequate emotion to circumstances or people is reduced.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 0.5 (0.6) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 0.4 (0.7) | 0.2 (0.5) | 0.8 (0.8)
  Month 3; n=24, 22, 17 | 0.6 (0.9) | 0.6 (0.9) | 0.6 (1.1)
  Month 6; n=25, 21, 17 | 0.6 (1.0) | 0.4 (0.7) | 0.8 (1.3)
  Month 9; n=25, 20, 17 | 0.5 (0.8) | 0.6 (0.6) | 0.7 (1.1)
  Month 12; n=25, 20, 17 | 0.6 (0.8) | 0.4 (0.6) | 0.5 (1.1)
  Month 18; n=24, 19, 16 | 0.5 (0.8) | 0.5 (0.6) | 0.8 (1.0)
  Month 24; n=23, 18, 15 | 0.5 (0.7) | 0.6 (0.7) | 1.1 (1.4)
  Month 30; n=23, 17, 13 | 0.4 (0.6) | 0.7 (0.7) | 0.7 (0.9)
  Month 36; n=21, 16, 12 | 0.6 (0.8) | 0.5 (0.7) | 0.7 (1.4)
  Endpoint; n=27, 22, 17 | 0.6 (0.8) | 0.6 (0.7) | 0.9 (1.4)

28. Secondary Outcome: MADRS Pessimistic Thoughts Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Pessimistic Thoughts scores rate thoughts of guilt, inferiority, self-reproach, sinfulness, remorse and ruin.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 0.9 (1.1) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 1.0 (0.8) | 0.5 (0.9) | 0.6 (0.8)
  Month 3; n=24, 22, 17 | 0.7 (0.9) | 0.5 (1.0) | 0.8 (1.0)
  Month 6; n=25, 21, 17 | 0.9 (0.9) | 0.6 (0.7) | 0.6 (0.9)
  Month 9; n=25, 20, 17 | 0.8 (0.8) | 0.5 (0.5) | 0.9 (1.0)
  Month 12; n=25, 20, 17 | 0.9 (0.8) | 0.8 (0.8) | 1.0 (0.9)
  Month 18; n=24, 19, 16 | 1.0 (0.8) | 0.7 (0.9) | 0.8 (0.8)
  Month 24; n=23, 18, 15 | 1.0 (1.0) | 0.7 (0.8) | 1.1 (0.9)
  Month 30; n=22, 17, 13 | 1.2 (0.9) | 0.7 (0.7) | 0.9 (0.8)
  Month 36; n=21, 16, 12 | 1.0 (1.0) | 0.9 (0.8) | 1.0 (1.1)
  Endpoint; n=26, 22, 17 | 1.2 (1.1) | 0.9 (0.8) | 1.1 (1.2)

29. Secondary Outcome: MADRS Suicidal Thoughts Scores From Baseline to Month 36
Description: MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Suicidal Thoughts scores rate the feeling that life is not worth living, that a natural death would be welcome, suicidal thoughts, and preparations for suicide.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=26, 0, 0 | 0.4 (0.6) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 0.5 (1.0) | 0.2 (0.6) | 0.3 (0.7)
  Month 3; n=24, 22, 17 | 0.5 (1.1) | 0.0 (0.2) | 0.4 (0.6)
  Month 6; n=25, 21, 17 | 0.5 (1.0) | 0.1 (0.4) | 0.2 (0.4)
  Month 9; n=25, 20, 17 | 0.3 (0.7) | 0.0 (0.0) | 0.2 (0.4)
  Month 12; n=25, 20, 17 | 0.3 (0.7) | 0.3 (0.4) | 0.2 (0.7)
  Month 18; n=24, 19, 16 | 0.5 (0.9) | 0.3 (0.7) | 0.2 (0.4)
  Month 24; n=23, 18, 15 | 0.1 (0.3) | 0.2 (0.5) | 0.4 (0.8)
  Month 30; n=23, 17, 13 | 0.4 (0.8) | 0.1 (0.3) | 0.2 (0.4)
  Month 36; n=21, 16, 12 | 0.5 (1.0) | 0.1 (0.3) | 0.1 (0.3)
  Endpoint; n=27, 22, 17 | 0.4 (0.9) | 0.2 (0.4) | 0.4 (0.8)

30. Secondary Outcome: Parkinson's Disease Questionnaire-39 (PDQ-39) Summary Index Scores From Baseline to Month 36
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. These include: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. The PDQ-39 Summary Index is the sum of all answers divided by the highest score possible, which is multiplied by 100 to put the score on a 0-100 scale. Higher scores are associated with more severe symptoms.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 33.6 (10.8) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 20, 17 | 27.1 (11.8) | 30.3 (10.7) | 36.6 (15.4)
  Month 3; n=22, 20, 18 | 24.5 (10.1) | 30.0 (15.6) | 34.0 (15.2)
  Month 6; n=24, 20, 17 | 27.9 (10.6) | 33.4 (16.2) | 35.5 (16.5)
  Month 9; n=23, 20, 16 | 25.9 (10.6) | 30.9 (12.1) | 35.1 (15.9)
  Month 12; n=23, 19, 17 | 28.8 (12.8) | 33.2 (15.5) | 38.3 (19.3)
  Month 18; n=22, 18, 16 | 28.2 (12.2) | 30.4 (15.7) | 34.1 (17.0)
  Month 24; n=21, 17, 14 | 30.3 (12.4) | 36.2 (14.6) | 33.6 (13.6)
  Month 30; n=21, 16, 12 | 33.5 (13.1) | 34.8 (16.2) | 34.4 (17.4)
  Month 36; n=20, 15, 11 | 36.8 (15.1) | 31.5 (11.5) | 39.2 (18.0)
  Endpoint; n=25, 21, 17 | 36.2 (14.1) | 34.0 (13.6) | 40.3 (17.5)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 0 (n=27); Test type: Superiority or Other; p = 0.001, Wilcoxon tests; mean change from baseline = -6.5, Standard Deviation 9.6
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 3 (n=23); Test type: Superiority or Other; p < 0.001, Wilcoxon tests; mean change from baseline = -9.2, Standard Deviation 9.0
Statistical Analysis 3: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 6 (n=24); Test type: Superiority or Other; p = 0.022, Wilcoxon tests; mean change from baseline = -5.9, Standard Deviation 11.2
Statistical Analysis 4: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 9 (n=23); Test type: Superiority or Other; p = 0.005, Wilcoxon tests; mean change from baseline = -7.5, Standard Deviation 11.6
Statistical Analysis 5: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 12 (n=23); Test type: Superiority or Other; p = 0.126, Wilcoxon tests; mean change from baseline = -5.3, Standard Deviation 13.9
Statistical Analysis 6: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 18 (n=22); Test type: Superiority or Other; p = 0.049, Wilcoxon tests; mean change from baseline = -5.2, Standard Deviation 12.3
Statistical Analysis 7: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 24 (n=21); Test type: Superiority or Other; p = 0.203, Wilcoxon tests; mean change from baseline = -3.1, Standard Deviation 9.9
Statistical Analysis 8: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 30 (n=21); Test type: Superiority or Other; p = 0.733, Wilcoxon tests; mean change from baseline = 0.8, Standard Deviation 13.2
Statistical Analysis 9: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Month 36 (n=20); Test type: Superiority or Other; p = 0.414, Wilcoxon tests; mean change from baseline = 4.4, Standard Deviation 14.3
Statistical Analysis 10: Comparison: Duodopa Naïve; Change from Baseline for the Duodopa Naïve group at Endpoint (n=27); Test type: Superiority or Other; p = 0.534, Wilcoxon tests; mean change from baseline = 2.3, Standard Deviation 14.9

31. Secondary Outcome: PDQ-39 Mobility Subscale Scores From Baseline to Month 36
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. These include: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 55.7 (20.5) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 38.8 (20.1) | 43.9 (21.7) | 53.3 (22.6)
  Month 3; n=23, 20, 18 | 36.0 (17.6) | 40.6 (22.8) | 50.6 (24.2)
  Month 6; n=25, 21, 18 | 39.5 (18.9) | 43.5 (23.5) | 54.7 (24.4)
  Month 9; n=24, 20, 17 | 40.2 (15.6) | 41.9 (21.7) | 52.8 (23.0)
  Month 12; n=25, 20, 17 | 41.0 (18.3) | 45.3 (24.2) | 54.4 (32.1)
  Month 18; n=24, 18, 16 | 40.9 (16.2) | 41.1 (25.6) | 54.7 (29.2)
  Month 24; n=21, 17, 15 | 46.0 (22.2) | 47.1 (21.5) | 49.5 (23.0)
  Month 30; n=22, 17, 12 | 50.9 (21.5) | 42.1 (21.5) | 53.3 (24.8)
  Month 36; n=21, 15, 11 | 57.3 (20.8) | 43.0 (21.6) | 61.1 (28.1)
  Endpoint; n=26, 21, 17 | 55.6 (20.7) | 50.2 (22.2) | 61.6 (25.0)

32. Secondary Outcome: PDQ-39 Activities of Daily Living Subscale Scores From Baseline to Month 36
Description: as for outcome 31
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 38.7 (21.5) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 20, 18 | 32.1 (19.0) | 40.8 (19.1) | 46.5 (26.5)
  Month 3; n=24, 22, 18 | 26.9 (16.6) | 42.8 (21.8) | 41.7 (22.2)
  Month 6; n=25, 21, 18 | 31.8 (18.9) | 43.7 (23.2) | 42.1 (22.5)
  Month 9; n=25, 20, 17 | 29.8 (19.2) | 37.5 (18.4) | 42.2 (21.3)
  Month 12; n=25, 20, 17 | 34.7 (20.8) | 42.1 (20.7) | 45.6 (26.5)
  Month 18; n=24, 20, 16 | 33.2 (20.1) | 41.9 (22.9) | 45.8 (24.6)
  Month 24; n=21, 17, 15 | 37.1 (22.1) | 48.3 (20.8) | 41.9 (24.1)
  Month 30; n=22, 17, 12 | 38.8 (23.8) | 48.5 (19.7) | 46.5 (28.2)
  Month 36; n=21, 15, 11 | 45.4 (25.1) | 47.5 (18.4) | 54.5 (29.3)
  Endpoint; n=26, 22, 17 | 43.4 (23.3) | 48.3 (18.2) | 53.4 (24.5)

33. Secondary Outcome: PDQ-39 Emotional Well Being Subscale Scores From Baseline to Month 36
Description: as for outcome 31
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 35.3 (19.3) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 30.9 (17.3) | 27.1 (19.3) | 37.7 (17.0)
  Month 3; n=23, 22, 18 | 24.8 (19.5) | 27.5 (19.6) | 35.4 (21.5)
  Month 6; n=25, 20, 18 | 31.3 (15.2) | 33.3 (18.6) | 35.9 (20.0)
  Month 9; n=25, 20, 17 | 33.0 (18.0) | 32.1 (17.0) | 34.8 (18.6)
  Month 12; n=25, 20, 17 | 29.0 (17.8) | 34.8 (20.8) | 38.0 (23.6)
  Month 18; n=24, 20, 16 | 32.1 (16.2) | 30.2 (19.5) | 32.6 (22.5)
  Month 24; n=21, 17, 15 | 31.9 (17.3) | 37.7 (19.0) | 33.1 (16.6)
  Month 30; n=22, 16, 12 | 33.9 (16.8) | 33.3 (25.2) | 31.3 (18.2)
  Month 36; n=21, 15, 11 | 39.7 (18.5) | 30.0 (21.0) | 38.6 (19.4)
  Endpoint; n=26, 22, 17 | 39.4 (17.8) | 31.1 (24.4) | 39.7 (21.5)

34. Secondary Outcome: PDQ-39 Stigma Subscale Scores From Baseline to Month 36
Description: as for outcome 31
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 24.8 (15.4) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 16.2 (16.8) | 16.5 (18.5) | 22.9 (23.0)
  Month 3; n=24, 22, 18 | 16.1 (15.0) | 18.8 (23.8) | 19.8 (17.4)
  Month 6; n=25, 21, 18 | 20.8 (16.2) | 19.0 (19.3) | 23.6 (24.4)
  Month 9; n=25, 20, 17 | 15.5 (15.7) | 12.8 (15.1) | 24.6 (23.6)
  Month 12; n=25, 19, 17 | 17.8 (17.0) | 19.4 (19.9) | 25.4 (25.5)
  Month 18; n=24, 20, 16 | 15.6 (17.5) | 13.8 (15.1) | 18.8 (22.0)
  Month 24; n=21, 17, 15 | 15.8 (12.4) | 23.5 (19.2) | 15.4 (14.5)
  Month 30; n=21, 17, 12 | 16.4 (18.6) | 14.0 (23.6) | 18.2 (21.4)
  Month 36; n=21, 15, 11 | 20.5 (19.1) | 12.9 (20.0) | 24.4 (19.3)
  Endpoint; n=26, 22, 17 | 19.5 (18.8) | 15.6 (20.3) | 25.0 (23.8)

35. Secondary Outcome: PDQ-39 Social Support Subscale Scores From Baseline to Month 36
Description: as for outcome 31
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27,0,0 | 8.3 (15.9) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 17 | 10.3 (18.2) | 12.9 (14.5) | 22.1 (19.1)
  Month 3; n=24, 22, 18 | 10.8 (15.2) | 12.5 (18.7) | 16.7 (19.6)
  Month 6; n=25, 21, 17 | 12.7 (18.0) | 13.1 (14.1) | 24.3 (21.5)
  Month 9; n=24, 20, 16 | 10.2 (16.3) | 13.8 (14.9) | 25.5 (18.1)
  Month 12; n=23, 20, 17 | 12.1 (19.5) | 19.6 (19.4) | 28.4 (22.6)
  Month 18; n=22, 20, 16 | 12.7 (15.6) | 17.9 (19.4) | 18.8 (18.4)
  Month 24; n=21, 17, 14 | 15.7 (18.5) | 20.6 (18.7) | 21.7 (15.7)
  Month 30; n=22, 17, 12 | 18.2 (24.8) | 16.2 (20.3) | 18.8 (22.8)
  Month 36; n=21, 15, 11 | 18.3 (21.0) | 11.7 (13.3) | 29.5 (26.7)
  Endpoint; n=26, 22, 17 | 21.8 (25.3) | 14.4 (18.9) | 27.9 (25.3)

36. Secondary Outcome: PDQ-39 Cognition Subscale Scores From Baseline to Month 36
Description: as for outcome 31
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 30.6 (15.6) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 22.5 (13.7) | 33.0 (16.6) | 33.7 (16.9)
  Month 3; n=24, 22, 18 | 24.2 (17.7) | 36.6 (18.5) | 32.3 (20.4)
  Month 6; n=24, 21, 18 | 25.5 (13.7) | 37.8 (18.3) | 30.6 (16.9)
  Month 9; n=25, 20, 17 | 21.5 (14.9) | 35.6 (20.0) | 31.6 (19.2)
  Month 12; n=25, 20, 17 | 26.8 (20.8) | 33.1 (19.7) | 33.8 (23.2)
  Month 18; n=24, 20, 16 | 28.6 (20.2) | 31.3 (22.1) | 30.1 (23.4)
  Month 24; n=21, 17, 15 | 24.7 (14.7) | 41.9 (16.8) | 27.5 (19.0)
  Month 30; n=22, 16, 12 | 31.5 (18.6) | 45.7 (23.7) | 30.7 (24.6)
  Month 36; n=20, 15, 11 | 34.1 (19.4) | 42.1 (16.6) | 30.7 (19.7)
  Endpoint; n=25, 22, 17 | 31.5 (19.8) | 39.2 (20.2) | 34.9 (19.5)

37. Secondary Outcome: PDQ-39 Communication Subscale Scores From Baseline to Month 36
Description: as for outcome 31
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 32.4 (21.6) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 24.1 (18.7) | 27.3 (14.6) | 35.2 (18.4)
  Month 3; n=24, 22, 18 | 24.7 (20.3) | 32.2 (22.2) | 31.9 (19.9)
  Month 6; n=24, 21, 18 | 24.0 (17.1) | 32.5 (22.0) | 33.8 (19.3)
  Month 9; n=25, 20, 17 | 25.3 (23.3) | 31.7 (17.2) | 28.9 (21.3)
  Month 12; n=25, 20, 17 | 29.7 (20.1) | 34.2 (18.3) | 33.8 (16.0)
  Month 18; n=24, 20, 16 | 31.6 (21.8) | 32.1 (19.0) | 29.7 (20.4)
  Month 24; n=21, 17, 15 | 28.2 (19.6) | 34.8 (18.2) | 30.6 (19.1)
  Month 30; n=22, 17, 12 | 33.7 (22.6) | 37.7 (18.4) | 41.7 (26.6)
  Month 36; n=21, 15, 11 | 33.7 (20.7) | 33.3 (13.0) | 37.9 (19.1)
  Endpoint; n=26, 22, 17 | 34.0 (20.9) | 33.0 (15.5) | 40.2 (18.7)

38. Secondary Outcome: PDQ-39 Bodily Discomfort Subscale Scores From Baseline to Month 36
Description: as for outcome 31
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Baseline (Month -3); n=27, 0, 0 | 42.6 (19.8) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Month 0; n=27, 22, 18 | 41.7 (18.3) | 40.2 (17.6) | 43.1 (24.8)
  Month 3; n=24, 22, 18 | 38.5 (21.7) | 39.8 (20.7) | 44.0 (21.4)
  Month 6; n=24, 21, 18 | 38.9 (22.1) | 42.1 (20.5) | 39.4 (23.2)
  Month 9; n=25, 20, 17 | 36.3 (18.8) | 42.1 (23.6) | 41.2 (24.7)
  Month 12; n=25, 20, 17 | 39.3 (21.0) | 34.6 (20.1) | 46.6 (27.6)
  Month 18; n=24, 20, 16 | 38.5 (23.5) | 37.1 (20.7) | 42.7 (24.5)
  Month 24; n=21, 17, 15 | 42.9 (24.2) | 35.3 (25.8) | 38.9 (23.7)
  Month 30; n=22, 17, 12 | 42.8 (23.3) | 39.2 (24.8) | 34.7 (27.3)
  Month 36; n=21, 15, 11 | 42.9 (17.9) | 31.7 (15.8) | 37.1 (20.2)
  Endpoint; n=26, 22, 17 | 42.6 (19.2) | 36.7 (20.5) | 39.7 (24.6)

39. Secondary Outcome: Electronic Diary: Morning and Day Scores (Walking) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. Walking scores ranged from 1 (worst) to 5 (best).
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Morning, Baseline (Month -3); n=20, 0, 0 | 2.7 (1.2) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 3.1 (0.9) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 3.3 (1.4) | 3.2 (1.1) | 3.4 (1.0)
  Day, Month 0; n=19, 20, 15 | 3.7 (1.1) | 3.7 (0.8) | 3.3 (1.0)
  Morning, Month 3; n=19, 19, 13 | 3.5 (1.1) | 3.0 (1.1) | 3.1 (1.0)
  Day, Month 3; n=19, 19, 13 | 3.7 (0.8) | 3.6 (1.0) | 3.3 (0.9)
  Morning, Month 6; n=16, 19, 11 | 3.5 (1.2) | 3.2 (1.1) | 3.3 (1.1)
  Day, Month 6; n=16, 19, 11 | 4.0 (0.7) | 3.7 (0.9) | 3.4 (0.9)
  Morning, Month 9; n=16, 17, 9 | 3.6 (1.0) | 3.3 (1.0) | 3.1 (1.3)
  Day, Month 9; n=16, 17, 9 | 4.0 (0.4) | 3.8 (0.9) | 3.1 (1.2)
  Morning, Month 12; n=16, 16, 9 | 3.6 (1.2) | 3.5 (1.1) | 3.1 (1.3)
  Day, Month 12; n=16, 16, 9 | 3.7 (1.0) | 3.8 (1.1) | 3.1 (1.2)
  Morning, Month 18; n=15, 14, 10 | 3.3 (1.2) | 3.5 (1.0) | 3.4 (1.1)
  Day, Month 18; n=15, 14, 10 | 3.8 (0.8) | 3.9 (0.8) | 3.5 (1.1)
  Morning, Month 24; n=14, 13, 7 | 3.4 (1.1) | 3.5 (1.0) | 2.9 (1.3)
  Day, Month 24; n=13, 13, 7 | 3.9 (0.4) | 3.9 (0.9) | 2.8 (1.5)
  Morning, Month 30; n=9, 9, 5 | 3.4 (1.3) | 3.4 (1.0) | 3.6 (0.9)
  Day, Month 30; n=9, 9, 5 | 3.8 (0.7) | 4.0 (0.5) | 3.9 (0.5)
  Morning, Month 36; n=6, 11, 5 | 2.3 (1.3) | 3.6 (1.0) | 3.7 (0.9)
  Day, Month 36; n=5, 11, 5 | 3.1 (1.3) | 4.0 (1.0) | 3.7 (0.6)
  Morning, Endpoint; n=23, 20, 16 | 2.8 (1.2) | 3.4 (1.0) | 3.0 (1.0)
  Day, Endpoint; n=23, 20, 16 | 3.4 (1.0) | 3.8 (0.9) | 3.0 (1.1)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.016, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.188, Wilcoxon tests

40. Secondary Outcome: Electronic Diary: Morning and Day Scores (Off Time) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. "Off" time is when PD symptoms are not adequately controlled by the drug, and is represented as a percentage of total time awake per day.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of 'off' time
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
percentage of 'off' time
  Morning, Baseline (Month -3); n=20, 0, 0 | 41.2 (19.4) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 35.4 (11.7) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 23.4 (19.7) | 30.6 (21.2) | 25.1 (12.7)
  Day, Month 0; n=19, 20, 15 | 20.8 (14.6) | 21.4 (9.2) | 25.7 (12.3)
  Morning, Month 3; n=19, 18, 13 | 26.4 (20.2) | 34.3 (20.0) | 25.7 (18.8)
  Day, Month 3; n=19, 19, 13 | 23.0 (12.8) | 22.7 (13.9) | 20.2 (10.3)
  Morning, Month 6; n=16, 19, 11 | 25.6 (21.0) | 30.1 (21.1) | 18.6 (10.9)
  Day, Month 6; n=16, 19, 11 | 21.9 (13.3) | 21.8 (15.3) | 20.9 (10.7)
  Morning, Month 9; n=16, 17, 9 | 23.9 (18.4) | 32.3 (20.5) | 23.6 (15.6)
  Day, Month 9; n=16, 17, 9 | 19.5 (13.4) | 21.5 (10.8) | 22.8 (11.6)
  Morning, Month 12; n=16, 16, 9 | 25.3 (17.8) | 28.0 (23.3) | 23.8 (16.0)
  Day, Month 12; n=16, 16, 9 | 24.0 (17.3) | 19.5 (16.0) | 23.5 (9.0)
  Morning, Month 18; n=15, 14, 10 | 21.1 (13.0) | 28.9 (21.4) | 24.9 (16.2)
  Day, Month 18; n=15, 14, 10 | 17.9 (8.6) | 21.6 (13.8) | 20.1 (11.9)
  Morning, Month 24; n=13, 13, 7 | 29.1 (21.6) | 25.4 (16.0) | 30.4 (17.9)
  Day, Month 24; n=13, 13, 7 | 22.0 (15.5) | 21.3 (14.2) | 24.9 (12.2)
  Morning, Month 30; n=9, 9, 5 | 23.4 (19.8) | 29.4 (23.1) | 28.0 (16.8)
  Day, Month 30; n=9, 9, 5 | 21.6 (15.1) | 24.0 (13.4) | 23.0 (11.2)
  Morning, Month 36; n=6, 11, 5 | 35.1 (25.2) | 29.4 (23.3) | 31.5 (15.1)
  Day, Month 36; n=5, 11, 5 | 24.7 (19.4) | 18.8 (11.7) | 23.6 (12.2)
  Morning, Endpoint; n=23, 20, 16 | 30.7 (22.8) | 28.5 (21.4) | 27.1 (13.8)
  Day, Endpoint; n=23, 20, 16 | 24.8 (17.2) | 22.3 (14.2) | 25.9 (11.7)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.008, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.107, Wilcoxon tests

41. Secondary Outcome: Electronic Diary: Morning and Day Scores (On Time) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. "On" time is when PD symptoms are well controlled by the drug, and is represented as a percentage of total time of the last __ hours.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of 'on' time
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
percentage of 'on' time
  Morning, Baseline (Month -3); n=20, 0, 0 | 40.2 (16.7) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 40.3 (14.0) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 58.4 (28.0) | 49.8 (23.1) | 55.2 (27.1)
  Day, Month 0; n=19, 20, 15 | 61.8 (19.8) | 60.2 (14.8) | 46.5 (28.0)
  Morning, Month 3; n=19, 18, 13 | 61.6 (23.6) | 52.0 (22.8) | 49.8 (28.2)
  Day, Month 3; n=19, 19, 13 | 62.6 (17.8) | 58.3 (20.7) | 55.0 (26.4)
  Morning, Month 6; n=16, 19, 11 | 57.7 (28.4) | 55.5 (24.1) | 55.8 (31.1)
  Day, Month 6; n=16, 19, 11 | 62.2 (22.0) | 57.3 (21.3) | 53.2 (29.7)
  Morning, Month 9; n=16, 17, 9 | 60.5 (25.1) | 52.3 (25.4) | 47.9 (29.4)
  Day, Month 9; n=16, 17, 9 | 59.7 (23.4) | 59.5 (18.1) | 50.8 (29.2)
  Morning, Month 12; n=16, 16, 9 | 61.1 (23.5) | 57.5 (23.4) | 49.0 (32.2)
  Day, Month 12; n=16, 16, 9 | 59.5 (25.0) | 63.0 (21.9) | 51.4 (26.9)
  Morning, Month 18; n=15, 14, 10 | 61.9 (21.4) | 55.2 (27.1) | 51.1 (33.4)
  Day, Month 18; n=15, 14, 10 | 61.5 (17.9) | 57.6 (20.7) | 52.5 (31.3)
  Morning, Month 24; n=13, 13, 7 | 61.3 (25.8) | 59.5 (23.1) | 41.3 (22.0)
  Day, Month 24; n=13, 13, 7 | 62.3 (21.7) | 57.4 (23.8) | 42.7 (24.8)
  Morning, Month 30; n=9, 9, 5 | 64.8 (28.3) | 49.3 (27.5) | 58.6 (26.3)
  Day, Month 30; n=9, 9, 5 | 62.4 (27.3) | 56.9 (20.1) | 58.8 (26.6)
  Morning, Month 36; n=6, 11, 5 | 54.5 (16.8) | 55.3 (23.4) | 51.9 (26.8)
  Day, Month 36; n=5, 11, 5 | 59.1 (14.8) | 61.8 (18.8) | 55.1 (28.2)
  Morning, Endpoint; n=23, 20, 16 | 52.9 (26.2) | 54.6 (21.8) | 49.9 (23.5)
  Day, Endpoint; n=23, 20, 16 | 56.0 (21.2) | 56.5 (18.0) | 46.2 (25.7)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.002, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.010, Wilcoxon tests

42. Secondary Outcome: Electronic Diary: Morning and Day Scores (Dyskinetic Time) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. 'Dyskinetic time' is time with involuntary muscle movement, and is represented as a percentage of total time of the last __ hours.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of 'dyskinetic' time
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
percentage of 'dyskinetic' time
  Morning, Baseline (Month -3); n=20, 0, 0 | 18.6 (12.4) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 24.3 (14.4) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 18.2 (24.2) | 19.6 (17.8) | 19.7 (17.5)
  Day, Month 0; n=19, 20, 15 | 17.4 (14.5) | 18.4 (12.5) | 27.3 (19.7)
  Morning, Month 3; n=19, 18, 13 | 12.0 (12.0) | 13.7 (13.6) | 24.5 (20.0)
  Day, Month 3; n=19, 19, 13 | 14.4 (13.0) | 18.9 (16.5) | 24.8 (21.3)
  Morning, Month 6; n=16, 19, 11 | 16.7 (17.3) | 14.4 (12.9) | 25.6 (24.3)
  Day, Month 6; n=16, 19, 11 | 15.9 (15.4) | 20.8 (16.3) | 25.8 (22.9)
  Morning, Month 9; n=16, 17, 9 | 15.6 (13.9) | 15.5 (9.4) | 28.5 (28.0)
  Day, Month 9; n=16, 17, 9 | 20.8 (15.4) | 19.0 (12.0) | 26.5 (22.8)
  Morning, Month 12; n=16, 16, 9 | 13.6 (13.2) | 14.6 (10.4) | 27.2 (24.8)
  Day, Month 12; n=16, 16, 9 | 16.2 (13.5) | 17.4 (13.8) | 25.1 (21.1)
  Morning, Month 18; n=15, 14, 10 | 17.0 (14.5) | 15.9 (11.6) | 24.0 (22.6)
  Day, Month 18; n=15, 14, 10 | 20.6 (11.9) | 20.8 (11.0) | 27.4 (21.2)
  Morning, Month 24; n=13, 13, 7 | 9.6 (12.0) | 15.0 (11.9) | 28.2 (19.5)
  Day, Month 24; n=13, 13, 7 | 15.8 (12.7) | 21.3 (19.0) | 32.4 (17.6)
  Morning, Month 30; n=9, 9, 5 | 11.8 (20.2) | 21.3 (15.2) | 13.4 (14.8)
  Day, Month 30; n=9, 9, 5 | 14.5 (16.8) | 19.1 (12.1) | 18.2 (16.9)
  Morning, Month 36; n=6, 11, 5 | 10.4 (9.8) | 15.2 (10.3) | 16.6 (18.0)
  Day, Month 36; n=5, 11, 5 | 16.2 (9.3) | 19.4 (10.8) | 21.3 (21.1)
  Morning, Endpoint; n=23, 20, 16 | 16.5 (21.4) | 16.9 (11.6) | 23.0 (15.5)
  Day, Endpoint; n=23, 20, 16 | 16.2 (9.3) | 19.4 (10.8) | 21.3 (21.1)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.048, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.003, Wilcoxon tests

43. Secondary Outcome: Electronic Diary: Morning and Day Scores (Off Magnitude) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. 'Off time' is when PD symptoms are not adequately controlled by the drug. Magnitude scores were 1 (worst) to 5 (best).
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Morning, Baseline (Month -3); n=20, 0, 0 | 2.7 (0.8) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 2.8 (0.5) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 3.6 (0.9) | 3.2 (0.9) | 3.4 (0.7)
  Day, Month 0; n=19, 20, 15 | 3.6 (0.7) | 3.5 (0.6) | 3.3 (0.6)
  Morning, Month 3; n=19, 18, 13 | 3.5 (0.8) | 2.8 (0.9) | 3.1 (0.9)
  Day, Month 3; 19, 19, 13 | 3.6 (0.5) | 3.6 (0.7) | 3.3 (0.6)
  Morning, Month 6; n=16, 19, 11 | 3.4 (0.9) | 3.2 (0.9) | 3.7 (0.6)
  Day, Month 6; 16, 19, 11 | 3.8 (0.5) | 3.7 (0.6) | 3.4 (0.6)
  Morning, Month 9; n=16, 17, 9 | 3.7 (0.8) | 3.3 (0.8) | 3.3 (0.5)
  Day, Month 9; n=16, 17, 9 | 3.8 (0.5) | 3.6 (0.7) | 3.2 (0.6)
  Morning, Month 12; n=16, 16, 9 | 3.7 (0.8) | 3.3 (1.0) | 3.4 (0.6)
  Day, Month 12; n=16, 16, 9 | 3.6 (0.7) | 3.6 (0.9) | 3.4 (0.6)
  Morning, Month 18; n=15, 14, 10 | 3.7 (0.7) | 3.3 (1.0) | 3.2 (0.7)
  Day, Month 18; n=15, 14, 10 | 3.8 (0.6) | 3.7 (0.7) | 3.5 (0.7)
  Morning, Month 24; n=13, 13, 7 | 3.6 (0.9) | 3.5 (0.8) | 3.1 (0.6)
  Day, Month 24; n=13, 13, 7 | 3.7 (0.7) | 3.6 (0.7) | 3.4 (0.6)
  Morning, Month 30; n=9, 9, 5 | 3.8 (0.9) | 3.3 (0.9) | 2.9 (0.7)
  Day, Month 30; n=9, 9, 5 | 3.8 (0.8) | 3.6 (0.7) | 3.2 (0.6)
  Morning, Month 36; n=6, 11, 5 | 3.1 (1.2) | 3.5 (0.8) | 3.2 (0.4)
  Day, Month 36; n=5, 11, 5 | 3.5 (0.8) | 3.8 (0.6) | 3.0 (0.8)
  Morning, Endpoint; n=23, 20, 16 | 3.3 (0.9) | 3.4 (0.8) | 3.3 (0.8)
  Day, Endpoint; n=23, 20, 16 | 3.5 (0.7) | 3.6 (0.6) | 3.1 (0.7)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.001, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.003, Wilcoxon tests

44. Secondary Outcome: Electronic Diary: Morning and Day Scores (Dyskinetic Magnitude) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. 'Dyskinetic time' is time with involuntary muscle movement. Magnitude scores were 1 (worst) to 5 (best).
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Morning, Baseline (Month -3); n=20, 0, 0 | 4.1 (0.8) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 3.6 (0.7) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 4.1 (0.8) | 4.1 (0.8) | 4.0 (0.6)
  Day, Month 0; n=19, 20, 15 | 4.0 (0.7) | 4.0 (0.5) | 3.7 (0.8)
  Morning, Month 3; n=19, 18, 13 | 4.4 (0.6) | 4.2 (0.5) | 4.0 (0.7)
  Day, Month 3; n=19, 19, 13 | 4.2 (0.6) | 4.0 (0.6) | 3.7 (0.8)
  Morning, Month 6; n=16, 19, 11 | 4.1 (0.6) | 4.1 (0.8) | 3.9 (0.7)
  Day, Month 6; n=16, 19, 11 | 4.2 (0.6) | 3.8 (0.8) | 3.7 (0.8)
  Morning, Month 9; n=16, 17, 9 | 4.1 (0.7) | 4.2 (0.6) | 3.7 (0.8)
  Day, Month 9; n=16, 17, 9 | 3.8 (0.7) | 4.0 (0.6) | 3.8 (0.6)
  Morning, Month 12; n=16, 16, 9 | 4.1 (0.6) | 4.2 (0.6) | 3.7 (0.7)
  Day, Month 12; n=16, 16, 9 | 4.1 (0.6) | 3.7 (0.8) | 3.8 (0.7)
  Morning, Month 18; n=15, 14, 10 | 3.9 (0.6) | 3.8 (0.7) | 3.9 (0.7)
  Day, Month 18; n=15, 14, 10 | 3.9 (0.5) | 3.9 (0.4) | 3.8 (0.8)
  Morning, Month 24; n=13, 13, 7 | 4.4 (0.6) | 4.2 (0.6) | 4.1 (0.6)
  Day, Month 24; n=13, 13, 7 | 4.1 (0.6) | 3.9 (0.6) | 3.8 (0.5)
  Morning, Month 30; n=9, 9, 5 | 4.5 (0.7) | 3.9 (0.6) | 4.2 (0.7)
  Day, Month 30; n=9, 9, 5 | 4.5 (0.5) | 3.9 (0.6) | 4.1 (0.6)
  Morning, Month 36; n=6, 11, 5 | 4.3 (0.8) | 4.0 (0.7) | 4.1 (0.6)
  Day, Month 36; n=5, 11, 5 | 4.0 (0.5) | 3.7 (0.6) | 4.0 (0.7)
  Morning, Endpoint; n=23, 20, 16 | 4.3 (0.8) | 4.0 (0.7) | 4.1 (0.6)
  Day, Endpoint; 23, 20, 16 | 4.0 (0.7) | 3.7 (0.6) | 3.6 (0.8)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 1.000, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.002, Wilcoxon tests

45. Secondary Outcome: Electronic Diary: Morning and Day Scores (Cramps) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. 'Cramps' scores were 1 (worst) to 5 (best).
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Morning, Baseline (Month -3); n=20, 0, 0 | 4.4 (0.7) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 4.5 (0.6) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 4.7 (0.4) | 4.6 (0.7) | 4.6 (0.4)
  Day, Month 0; n=19, 20, 15 | 4.7 (0.4) | 4.7 (0.5) | 4.6 (0.5)
  Morning, Month 3; n=19, 18, 13 | 4.8 (0.3) | 4.6 (0.7) | 4.5 (0.6)
  Day, Month 3; n=19, 19, 13 | 4.7 (0.5) | 4.7 (0.6) | 4.5 (0.7)
  Morning, Month 6; n=16, 19, 11 | 4.8 (0.3) | 4.5 (0.9) | 4.3 (1.2)
  Day, Month 6; n=16, 19, 11 | 4.8 (0.3) | 4.5 (0.8) | 4.3 (1.1)
  Morning, Month 9; n=16, 17, 9 | 4.8 (0.3) | 4.4 (0.7) | 4.4 (1.0)
  Day, Month 9; n=16, 17, 9 | 4.7 (0.5) | 4.5 (0.7) | 4.3 (0.9)
  Morning, Month 12; n=16, 16, 9 | 4.8 (0.3) | 4.5 (0.7) | 4.2 (1.4)
  Day, Month 12; n=16, 16, 9 | 4.5 (0.7) | 4.7 (0.5) | 4.1 (1.3)
  Morning, Month 18; n=15, 14, 10 | 4.7 (0.4) | 4.4 (0.8) | 4.1 (0.8)
  Day, Month 18; n=15, 14, 10 | 4.7 (0.5) | 4.6 (0.5) | 4.3 (1.0)
  Morning, Month 24; n=13, 13, 7 | 4.6 (0.4) | 4.8 (0.2) | 4.0 (1.4)
  Day, Month 24; n=13, 13, 7 | 4.5 (0.6) | 4.8 (0.3) | 4.0 (1.3)
  Morning, Month 30; n=9, 9, 5 | 4.9 (0.3) | 4.7 (0.4) | 4.1 (1.5)
  Day, Month 30; n=9, 9, 5 | 4.9 (0.3) | 4.8 (0.2) | 3.9 (1.5)
  Morning, Month 36; n=6, 11, 5 | 4.5 (0.4) | 4.7 (0.3) | 4.1 (1.3)
  Day, Month 36; n=5, 11, 5 | 4.7 (0.6) | 4.8 (0.2) | 4.2 (1.0)
  Morning, Endpoint; n=23, 20, 16 | 4.6 (0.4) | 4.5 (0.7) | 4.4 (0.8)
  Day, Endpoint; n=23, 20, 16 | 4.5 (0.6) | 4.6 (0.5) | 4.5 (0.7)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.017, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Test type: Superiority or Other; p = 0.191, Wilcoxon tests

46. Secondary Outcome: Electronic Diary: Morning and Day Scores (Satisfied With Function) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. 'Satisfied with function' scores were 1 (worst) to 5 (best).
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Morning, Baseline (Month -3); n=20, 0, 0 | 2.5 (1.0) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 2.6 (0.5) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 3.3 (0.9) | 3.2 (0.9) | 3.8 (0.8)
  Day, Month 0; n=19, 20, 15 | 3.4 (0.7) | 3.4 (0.6) | 3.3 (1.0)
  Morning, Month 3; n=19, 18, 13 | 3.4 (0.9) | 3.0 (1.1) | 3.4 (1.1)
  Day, Month 3; n=19, 19, 13 | 3.5 (0.6) | 3.4 (0.8) | 3.3 (0.9)
  Morning, Month 6; n=16, 19, 11 | 3.5 (0.9) | 3.3 (0.8) | 3.7 (0.8)
  Day, Month 6; n=16, 19, 11 | 3.6 (0.6) | 3.4 (0.7) | 3.5 (0.7)
  Morning, Month 9; n=16, 17, 9 | 3.4 (0.7) | 3.3 (0.9) | 3.6 (0.7)
  Day, Month 9; n=16, 17, 9 | 3.5 (0.6) | 3.4 (0.8) | 3.4 (0.7)
  Morning, Month 12; n=16, 16, 9 | 3.6 (0.8) | 3.4 (0.8) | 3.5 (0.8)
  Day, Month 12; n=16, 16, 9 | 3.5 (0.6) | 3.6 (0.6) | 3.6 (0.7)
  Morning, Month 18; n=15, 14, 10 | 3.4 (0.9) | 3.4 (0.8) | 3.3 (1.1)
  Day, Month 18; n=15, 14, 10 | 3.5 (0.6) | 3.6 (0.5) | 3.4 (0.8)
  Morning, Month 24; n=13, 13, 7 | 3.4 (0.9) | 3.6 (0.7) | 3.1 (0.9)
  Day, Month 24; n=13, 13, 7 | 3.6 (0.6) | 3.5 (0.7) | 3.3 (0.9)
  Morning, Month 30; n=9, 9, 5 | 3.6 (0.8) | 3.4 (0.9) | 3.6 (0.9)
  Day, Month 30; n=9, 9, 5 | 3.5 (0.8) | 3.6 (0.5) | 3.6 (0.5)
  Morning, Month 36; n=6, 11, 5 | 3.4 (0.4) | 3.3 (0.8) | 3.5 (0.9)
  Day, Month 36; n=5, 11, 5 | 3.5 (0.5) | 3.5 (0.7) | 3.5 (0.8)
  Morning, Endpoint; n=23, 20, 16 | 3.2 (0.7) | 3.3 (0.7) | 3.4 (0.9)
  Day, Endpoint; n=23, 20, 16 | 3.4 (0.6) | 3.4 (0.6) | 3.1 (0.9)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.002, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p < 0.001, Wilcoxon tests

47. Secondary Outcome: Electronic Diary: Morning and Day Scores (Self-assessment) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. 'Self-assessment' scores were -3 (Off) to +3 (dyskinetic). 'Off' time is when PD symptoms are not adequately controlled by the drug. 'Dyskinetic' time is time with involuntary muscle movement. "0" is defined as the normal ON state without dyskinesia (the desired motor state). Everything closer to "0" means improvement, everything more away from "0" means either less mobility (in the negative score) or involuntary movements (dyskinesia, in the positive score).
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Morning, Baseline (Month -3); n=20, 0, 0 | -0.9 (1.2) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | -0.3 (1.1) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | -0.4 (1.1) | -0.1 (1.0) | 0.2 (0.8)
  Day, Month 0; n=19, 20, 15 | -0.2 (0.9) | -0.1 (0.6) | 0.1 (1.0)
  Morning, Month 3; n=19, 18, 13 | -0.2 (0.9) | -0.6 (0.9) | 0.0 (0.8)
  Day, Month 3; n=19, 19, 13 | -0.3 (0.7) | -0.1 (0.7) | 0.3 (1.0)
  Morning, Month 6; n=16, 19, 11 | -0.4 (1.0) | -0.2 (1.0) | 0.3 (0.7)
  Day, Month 6; n=16, 19, 11 | -0.2 (0.8) | 0.0 (0.8) | 0.3 (0.7)
  Morning, Month 9; n=16, 17, 9 | -0.2 (0.8) | -0.4 (0.7) | 0.4 (1.0)
  Day, Month 9; n=16, 17, 9 | 0.2 (0.8) | -0.0 (0.5) | -0.1 (0.6)
  Morning, Month 12; n=16, 16, 9 | -0.3 (0.8) | -0.2 (0.9) | 0.4 (0.6)
  Day, Month 12; n=16, 16, 9 | -0.3 (0.9) | 0.1 (0.8) | 0.1 (0.8)
  Morning, Month 18; n=15, 14, 10 | -0.3 (0.8) | 0.1 (0.8) | -0.0 (0.9)
  Day, Month 18; n=15, 14, 10 | -0.2 (0.7) | -0.2 (0.4) | 0.1 (0.9)
  Morning, Month 24; n=13, 13, 7 | -0.5 (0.8) | -0.0 (0.7) | 0.1 (0.9)
  Day, Month 24; n=13, 13, 7 | -0.2 (0.8) | -0.1 (0.8) | -0.0 (0.5)
  Morning, Month 30; n=9, 9, 5 | -0.4 (1.2) | -0.2 (0.9) | 0.2 (1.1)
  Day, Month 30; n=9, 9, 5 | -0.3 (0.8) | -0.3 (0.5) | -0.3 (0.5)
  Morning, Month 36; n=6, 11, 5 | -0.9 (1.3) | -0.0 (1.2) | 0.3 (0.7)
  Day, Month 36; n=5, 11, 5 | -0.2 (1.0) | 0.2 (0.5) | -0.2 (0.8)
  Morning, Endpoint; n=23, 20, 16 | -0.6 (1.1) | -0.2 (1.1) | 0.2 (0.7)
  Day, Endpoint; n=23, 20, 16 | -0.3 (1.0) | -0.0 (0.7) | 0.2 (1.0)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.047, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.847, Wilcoxon tests

48. Secondary Outcome: Electronic Diary: Morning and Day Scores (Free Tapping - Speed) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. Free tapping is defined as voluntary repetitive finger tapping on computer-generated fields. 'Free tapping speed' is a count of the number of taps per 20 seconds.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: taps/20 seconds
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
taps/20 seconds
  Morning, Baseline (Month -3); n=20, 0, 0 | 39.9 (12.8) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 39.7 (11.2) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 44.4 (12.5) | 39.2 (14.2) | 40.6 (14.1)
  Day, Month 0; n=19, 20, 15 | 43.5 (11.5) | 40.2 (12.5) | 40.3 (13.0)
  Morning, Month 3; n=19, 18, 13 | 46.8 (15.1) | 42.2 (15.6) | 46.3 (13.6)
  Day, Month 3; n=19, 19, 13 | 47.4 (13.8) | 43.2 (14.5) | 43.2 (12.9)
  Morning, Month 6; n=16, 19, 11 | 50.7 (15.5) | 43.4 (17.5) | 48.0 (14.3)
  Day, Month 6; n=16, 19, 11 | 50.3 (14.9) | 43.0 (15.8) | 47.6 (12.0)
  Morning, Month 9; n=16, 17, 9 | 47.2 (13.3) | 45.7 (20.0) | 46.8 (16.0)
  Day, Month 9; n=16, 17, 9 | 48.1 (15.7) | 48.0 (16.8) | 47.0 (15.3)
  Morning, Month 12; n=16, 16, 9 | 49.3 (16.0) | 44.5 (16.1) | 47.0 (18.8)
  Day, Month 12; n=16, 16, 9 | 48.7 (17.6) | 46.6 (15.1) | 46.6 (18.5)
  Morning, Month 18; n=15, 14, 10 | 44.0 (14.1) | 43.1 (17.5) | 46.7 (18.9)
  Day, Month 18; n=15, 14, 10 | 46.9 (12.5) | 46.3 (15.1) | 45.9 (18.1)
  Morning, Month 24; n=13, 13, 7 | 47.3 (14.9) | 45.5 (17.6) | 38.7 (14.7)
  Day, Month 24; n=13, 13, 7 | 47.6 (15.0) | 48.7 (14.2) | 41.5 (12.9)
  Morning, Month 30; n=9, 9, 5 | 49.4 (15.7) | 42.2 (18.1) | 49.3 (22.5)
  Day, Month 30; n=9, 9, 5 | 49.5 (13.0) | 42.6 (16.1) | 52.6 (19.1)
  Morning, Month 36; n=6, 11, 5 | 46.3 (14.0) | 44.7 (18.6) | 51.4 (25.0)
  Day, Month 36; n=5, 11, 5 | 45.5 (8.5) | 45.6 (19.7) | 50.5 (23.6)
  Morning, Endpoint; n=23, 20, 16 | 41.8 (11.6) | 41.2 (16.8) | 43.1 (16.8)
  Day, Endpoint; n=23, 20, 16 | 43.6 (12.1) | 43.2 (16.6) | 41.4 (15.0)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.012, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.035, Wilcoxon tests

49. Secondary Outcome: Electronic Diary: Morning and Day Scores (Free Tapping - Accuracy) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. 'Free tapping' is defined as ____. 'Free tapping accuracy' is the percentage of accurate free taps per 20 seconds(?).
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of tapping accuracy
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
percentage of tapping accuracy
  Morning, Baseline (Month -3); n=20, 0, 0 | 70.7 (16.4) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 71.9 (14.2) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 71.4 (16.2) | 69.8 (13.8) | 63.8 (13.1)
  Day, Month 0; n=19, 20, 15 | 70.1 (14.6) | 70.7 (12.4) | 65.2 (10.1)
  Morning, Month 3; n=19, 18, 13 | 73.4 (13.0) | 70.3 (13.9) | 63.5 (13.4)
  Day, Month 3; n=19, 19, 13 | 70.0 (14.4) | 69.7 (12.4) | 65.8 (12.9)
  Morning, Month 6; n=16, 19, 11 | 67.6 (9.4) | 66.2 (13.8) | 64.8 (17.2)
  Day, Month 6; n=16, 19, 11 | 65.7 (13.0) | 66.1 (12.6) | 66.7 (14.1)
  Morning, Month 9; n=16, 17, 9 | 67.0 (13.3) | 63.6 (16.9) | 65.8 (14.2)
  Day, Month 9; n=16, 17, 9 | 65.4 (9.3) | 69.9 (13.4) | 67.5 (10.9)
  Morning, Month 12; n=16, 16, 9 | 68.7 (15.3) | 71.5 (14.4) | 61.5 (8.8)
  Day, Month 12; n=16, 16, 9 | 64.7 (16.9) | 71.7 (11.9) | 60.4 (9.1)
  Morning, Month 18; n=15, 14, 10 | 58.9 (10.8) | 65.4 (18.2) | 65.8 (13.3)
  Day, Month 18; n=15, 14, 10 | 61.2 (11.0) | 69.1 (12.3) | 61.4 (12.7)
  Morning, Month 24; n=13, 13, 7 | 62.3 (16.9) | 66.2 (16.7) | 61.9 (14.3)
  Day, Month 24; n=13, 13, 7 | 64.4 (14.5) | 69.1 (15.9) | 62.4 (11.7)
  Morning, Month 30; n=9, 9, 5 | 66.3 (10.6) | 67.2 (12.8) | 62.1 (13.6)
  Day, Month 30; n=9, 9, 5 | 66.8 (12.1) | 67.3 (12.3) | 67.9 (10.5)
  Morning, Month 36; n=6, 11, 5 | 60.7 (24.1) | 60.3 (19.3) | 61.2 (12.6)
  Day, Month 36; n=5, 11, 5 | 50.3 (13.0) | 64.6 (15.5) | 63.6 (11.2)
  Morning, Endpoint; n=23, 20, 16 | 63.7 (17.1) | 58.7 (17.0) | 59.3 (13.6)
  Day, Endpoint; n=23, 20, 16 | 60.1 (15.8) | 62.7 (14.7) | 60.3 (13.7)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.599, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.048, Wilcoxon tests

50. Secondary Outcome: Electronic Diary: Morning and Day Scores (Tapping, Increased Speed - Accuracy) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. 'Tapping at increased speed - accuracy' is the percentage of accurate taps per all taps on computer-generated fields.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of accurate taps
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
percentage of accurate taps
  Morning, Baseline (Month -3); n=20, 0, 0 | 74.6 (13.9) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 73.7 (14.7) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 83.7 (12.0) | 71.0 (24.8) | 73.2 (15.1)
  Day, Month 0; n=19, 20, 15 | 80.4 (10.6) | 73.9 (18.6) | 73.2 (13.8)
  Morning, Month 3; n=19, 18, 13 | 83.1 (14.8) | 73.5 (22.3) | 68.8 (22.7)
  Day, Month 3; n=19, 19, 13 | 81.3 (14.5) | 74.7 (20.5) | 69.3 (20.2)
  Morning, Month 6; n=16, 19, 11 | 87.1 (11.0) | 74.2 (22.1) | 73.3 (20.1)
  Day, Month 6; n=16, 19, 11 | 87.8 (9.8) | 73.6 (20.3) | 73.0 (21.2)
  Morning, Month 9; n=16, 17, 9 | 86.4 (11.1) | 78.2 (19.0) | 77.1 (16.9)
  Day, Month 9; n=16, 17, 9 | 86.0 (10.1) | 78.8 (15.3) | 75.6 (19.0)
  Morning, Month 12; n=16, 16, 9 | 87.0 (12.5) | 80.1 (18.6) | 74.6 (20.0)
  Day, Month 12; n=16, 16, 9 | 81.8 (15.6) | 77.5 (20.9) | 72.4 (23.6)
  Morning, Month 18; n=15, 14, 10 | 81.3 (13.9) | 77.9 (18.5) | 71.4 (25.8)
  Day, Month 18; n=15, 14, 10 | 82.1 (12.9) | 78.7 (19.2) | 72.1 (24.4)
  Morning, Month 24; n=13, 13, 7 | 85.7 (13.1) | 79.4 (20.6) | 69.0 (18.9)
  Day, Month 24; n=13, 13, 7 | 85.3 (10.6) | 82.0 (15.9) | 70.0 (16.9)
  Morning, Month 30; n=9, 9, 5 | 87.3 (5.1) | 73.5 (21.1) | 79.8 (18.1)
  Day, Month 30; n=9, 9, 5 | 88.6 (6.4) | 74.5 (19.7) | 80.6 (20.5)
  Morning, Month 36; n=6, 11, 5 | 77.9 (18.8) | 71.7 (24.9) | 81.0 (17.3)
  Day, Month 36; n=5, 11, 5 | 70.7 (15.9) | 72.8 (21.8) | 77.9 (21.1)
  Morning, Endpoint; n=23, 20, 16 | 79.5 (17.7) | 70.4 (23.8) | 68.0 (19.7)
  Day, Endpoint; n=23, 20, 16 | 74.6 (17.4) | 72.0 (22.2) | 67.5 (20.5)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.026, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.208, Wilcoxon tests

51. Secondary Outcome: Electronic Diary: Morning and Day Scores (Tapping, Random Chase - Speed) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. Tapping: Random chase speed' is defined as the number of correct taps of fields randomly selected by the computer per 20 seconds.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: taps/20 seconds
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
taps/20 seconds
  Morning, Baseline (Month -3); n=20, 0, 0 | 24.5 (4.1) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 24.2 (4.2) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 26.3 (4.8) | 22.6 (5.8) | 22.7 (4.7)
  Day, Month 0; n=19, 20, 15 | 26.3 (5.0) | 23.4 (5.4) | 22.0 (4.9)
  Morning, Month 3; n=19, 18, 13 | 27.2 (5.1) | 23.8 (5.9) | 24.3 (3.5)
  Day, Month 3; n=19, 19, 13 | 27.2 (4.7) | 24.4 (6.3) | 24.0 (3.9)
  Morning, Month 6; n=16, 19, 11 | 28.3 (4.7) | 24.2 (5.3) | 24.4 (4.1)
  Day, Month 6; n=16, 19, 11 | 28.2 (4.5) | 24.4 (5.3) | 25.3 (4.2)
  Morning, Month 9; n=16, 17, 9 | 27.2 (4.1) | 24.4 (5.4) | 25.0 (5.0)
  Day, Month 9; n=16, 17, 9 | 27.0 (4.5) | 25.6 (4.4) | 25.6 (4.7)
  Morning, Month 12; n=16, 16, 9 | 27.2 (5.4) | 25.5 (5.1) | 23.8 (5.4)
  Day, Month 12; n=16, 16, 9 | 26.3 (5.3) | 26.4 (4.9) | 24.7 (5.5)
  Morning, Month 18; n=15, 14, 10 | 26.2 (4.1) | 24.9 (6.4) | 24.8 (6.1)
  Day, Month 18; n=15, 14, 10 | 26.3 (3.7) | 25.9 (6.1) | 25.0 (7.0)
  Morning, Month 24; n=13, 13, 7 | 27.0 (5.2) | 24.8 (5.6) | 22.7 (5.1)
  Day, Month 24; n=13, 13, 7 | 26.7 (5.6) | 26.5 (5.1) | 23.8 (4.6)
  Morning, Month 30; n=9, 9, 5 | 27.4 (4.6) | 24.4 (6.1) | 25.1 (7.0)
  Day, Month 30; n=9, 9, 5 | 27.9 (4.2) | 25.1 (5.8) | 27.0 (5.3)
  Morning, Month 36; n=6, 11, 5 | 26.5 (5.3) | 23.1 (6.7) | 25.1 (6.8)
  Day, Month 36; n=5, 11, 5 | 25.2 (2.4) | 23.9 (6.3) | 26.3 (6.3)
  Morning, Endpoint; n=23, 20, 16 | 25.1 (5.5) | 22.7 (6.3) | 22.8 (5.2)
  Day, Endpoint; 23, 20, 16 | 25.1 (4.8) | 23.6 (6.2) | 23.0 (6.3)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.010, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.073, Wilcoxon tests

52. Secondary Outcome: Electronic Diary: Morning and Day Scores (Tapping, Random Chase - Accuracy) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. Tapping: Random chase speed' is defined as the number of correct taps of fields randomly selected by the computer per 20 seconds. 'Tapping random chase - accuracy' is the percentage of accurate random chase taps.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of accurate taps
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
percentage of accurate taps
  Morning, Baseline (Month -3); n=20, 0, 0 | 92.0 (14.2) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 91.8 (7.8) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 94.6 (4.5) | 90.0 (12.6) | 92.6 (6.3)
  Day, Month 0; n=19, 20, 15 | 92.9 (6.8) | 91.3 (10.6) | 92.3 (7.0)
  Morning, Month 3; n=19, 18, 13 | 90.5 (17.3) | 89.2 (11.6) | 89.1 (10.1)
  Day, Month 3; n=19, 19, 13 | 92.5 (9.8) | 88.6 (13.6) | 89.8 (8.0)
  Morning, Month 6; n=16, 19, 11 | 95.2 (4.4) | 89.0 (14.2) | 90.5 (7.7)
  Day, Month 6; n=16, 19, 11 | 94.6 (3.5) | 88.7 (14.0) | 89.2 (11.6)
  Morning, Month 9; n=16, 17, 9 | 91.2 (8.1) | 90.8 (10.5) | 91.8 (6.3)
  Day, Month 9; n=16, 17, 9 | 92.4 (7.7) | 93.1 (7.2) | 92.5 (4.8)
  Morning, Month 12; n=16, 16, 9 | 92.2 (8.8) | 90.7 (11.4) | 90.6 (5.9)
  Day, Month 12; n=16, 16, 9 | 91.2 (7.6) | 92.5 (8.0) | 89.2 (7.9)
  Morning, Month 18; n=15, 14, 10 | 90.2 (11.3) | 88.8 (14.6) | 86.8 (13.9)
  Day, Month 18; n=15, 14, 10 | 91.6 (5.5) | 92.1 (9.2) | 85.4 (15.4)
  Morning, Month 24; n=13, 13, 7 | 91.7 (10.2) | 92.2 (9.6) | 89.0 (7.7)
  Day, Month 24; n=13, 13, 7 | 92.9 (6.7) | 93.4 (5.2) | 90.7 (6.3)
  Morning, Month 30; n=9, 9, 5 | 95.1 (3.3) | 85.9 (11.5) | 90.5 (9.1)
  Day, Month 30; n=9, 9, 5 | 93.6 (4.9) | 88.6 (8.6) | 91.2 (7.2)
  Morning, Month 36; n=6, 11, 5 | 83.5 (19.8) | 85.9 (14.8) | 89.7 (7.0)
  Day, Month 36; n=5, 11, 5 | 82.1 (16.9) | 88.4 (11.8) | 88.8 (7.5)
  Morning, Endpoint; n=23, 20, 16 | 87.8 (18.7) | 83.8 (15.1) | 87.5 (8.1)
  Day, Endpoint; n=23, 20, 16 | 87.3 (12.6) | 86.6 (14.3) | 86.7 (9.6)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.048, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.030, Wilcoxon tests

53. Secondary Outcome: Electronic Diary: Morning and Day Scores (Drawing Impairment [Wavelet Method]) From Baseline to Month 36
Description: The Electronic Diary consisted of 15 items addressing motor performance, complication of therapy, self-assessment, and various types of tapping. Six conceptual dimensions were defined; four subjectively-reported: 'walking', 'satisfied', 'dyskinesia', and 'off' and two objectively-measured: 'tapping' and 'spiral'. Each of the items was assessed in the morning and during the day. Drawing impairment was assessed as a spiral score, where the participant is asked to draw a spiral. 1 is worst score, 10 is best.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Morning, Baseline (Month -3); n=20, 0, 0 | 4.0 (1.4) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Day, Baseline (Month -3); n=20, 0, 0 | 4.0 (1.2) | NA (NA) — Baseline for Duodopa non-naive participants was not done. | NA (NA) — Baseline for Duodopa non-naive participants was not done.
  Morning, Month 0; n=19, 20, 15 | 4.1 (1.4) | 4.5 (1.6) | 5.0 (1.2)
  Day, Month 0; n=19, 20, 15 | 4.2 (1.3) | 4.3 (1.5) | 5.1 (1.2)
  Morning, Month 3; n=19, 18, 13 | 3.6 (1.2) | 4.3 (1.5) | 4.7 (1.5)
  Day, Month 3; n=19, 19, 13 | 3.8 (1.2) | 4.2 (1.4) | 4.8 (1.5)
  Morning, Month 6; n=16, 19, 11 | 3.8 (1.3) | 4.5 (1.7) | 4.5 (1.4)
  Day, Month 6; n=16, 19, 11 | 4.1 (1.0) | 4.6 (1.6) | 4.5 (1.7)
  Morning, Month 9; n=16, 17, 9 | 4.3 (1.2) | 4.1 (1.4) | 4.6 (1.5)
  Day, Month 9; n=16, 17, 9 | 4.3 (1.0) | 4.1 (1.2) | 4.5 (1.5)
  Morning, Month 12; n=16, 16, 9 | 4.1 (1.5) | 4.1 (1.2) | 5.0 (1.4)
  Day, Month 12; n=16, 16, 9 | 4.4 (1.2) | 4.1 (1.3) | 4.7 (1.4)
  Morning, Month 18; n=15, 14, 10 | 4.6 (1.3) | 4.4 (1.5) | 5.4 (1.8)
  Day, Month 18; n=15, 14, 10 | 4.6 (1.0) | 4.3 (1.5) | 4.9 (1.8)
  Morning, Month 24; n=13, 13, 7 | 4.3 (1.5) | 3.9 (1.3) | 5.2 (1.7)
  Day, Month 24; n=13, 13, 7 | 4.5 (1.4) | 3.9 (1.1) | 5.1 (1.7)
  Morning, Month 30; n=9, 9, 5 | 4.1 (1.4) | 4.4 (1.5) | 4.9 (1.5)
  Day, Month 30; n=9, 9, 5 | 4.5 (1.2) | 4.4 (1.4) | 4.8 (1.9)
  Morning, Month 36; n=6, 11, 5 | 4.4 (1.6) | 4.8 (1.8) | 5.3 (1.6)
  Day, Month 36; n=5, 11, 5 | 5.0 (0.9) | 4.6 (1.5) | 5.3 (1.3)
  Morning, Endpoint; n=23, 20, 16 | 4.5 (1.4) | 5.0 (1.8) | 5.3 (1.3)
  Day, Endpoint; n=23, 20, 16 | 4.8 (1.2) | 4.9 (1.7) | 5.3 (1.2)
Statistical Analysis 1: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for morning scores; Test type: Superiority or Other; p = 0.208, Wilcoxon tests
Statistical Analysis 2: Comparison: Duodopa Naïve; Change from Baseline to Month 12 for day scores; Test type: Superiority or Other; p = 0.048, Wilcoxon tests

54. Other Pre Specified Outcome: UPDRS Total Score up to Month 36
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. For Parts I-III and Total Score, each question is measured on a 5-point scale of 0 (normal or no disease effect) to 4 (maximum negative effect). Part I score is the sum of answers to 'Mentation, Behavior and Mood' questions, with a score range from 0-16. Part II score is the sum of answers to 'Activities of Daily Living' questions, with a score range from 0-52. Part III score is the sum of answers to 'Motor Examination' questions, with a score range from 0-108. Total Score is the sum of the responses to the 31 questions (44 answers) that comprise Parts I-III of the scale, with a score range from 0-176. Higher scores are associated with more disability.
Time Frame: Months 0, 3, 6, 9, 18, 24, 30, 36, endpoint (last non-missing value assigned to treatment for the participant)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Month 0; n=27, 22, 18 | 43.1 (16.7) | 46.2 (17.3) | 47.8 (16.4)
  Month 3; n=24, 22, 18 | 42.4 (19.1) | 45.5 (18.2) | 46.8 (16.4)
  Month 6; n=25, 22, 18 | 43.3 (21.4) | 43.5 (17.6) | 47.4 (13.2)
  Month 9; 5, 20, 17 | 40.8 (22.4) | 45.1 (13.0) | 48.1 (17.8)
  Month 18; n=24, 20, 17 | 45.2 (22.8) | 44.2 (16.1) | 48.5 (18.0)
  Month 24; n=23, 18, 15 | 44.5 (25.3) | 40.2 (15.9) | 52.7 (15.5)
  Month 30; n=23, 17, 13 | 47.1 (25.5) | 47.4 (19.0) | 50.2 (19.8)
  Month 36; n=21, 16, 12 | 46.2 (27.8) | 47.1 (14.3) | 54.0 (25.3)
  Endpoint visit; n=27, 22, 18 | 47.9 (25.8) | 50.8 (17.5) | 55.0 (23.0)

55. Other Pre Specified Outcome: UPDRS Part I Score, up to Month 36
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. For Parts I-III and Total Score, each question is measured on a 5-point scale of 0 (normal or no disease effect) to 4 (maximum negative effect). Part I score is the sum of answers to 'Mentation, Behavior and Mood' questions, with a score range from 0-16. Higher scores are associated with more disability.
Time Frame: Months 0, 3, 6, 9, 18, 24, 30, 36, endpoint (last non-missing value assigned to treatment for the participant)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Month 0; n=27, 22, 18 | 2.4 (1.8) | 2.0 (1.8) | 2.7 (1.8)
  Month 3; n=24, 22, 18 | 2.5 (1.7) | 2.0 (1.6) | 3.2 (2.3)
  Month 6; n=25, 22, 18 | 2.9 (1.9) | 2.3 (1.8) | 2.9 (2.1)
  Month 9; n=25, 20, 17 | 3.0 (1.9) | 2.9 (1.6) | 3.3 (2.3)
  Month 18; n=24, 20, 17 | 4.1 (3.0) | 2.7 (2.2) | 3.3 (2.6)
  Month 24; n=23, 18, 15 | 3.9 (2.8) | 3.0 (2.0) | 3.5 (2.1)
  Month 30; n=23, 17, 13 | 4.1 (3.2) | 3.5 (2.7) | 2.8 (2.0)
  Month 36; n=21, 16, 12 | 3.9 (3.1) | 3.9 (2.5) | 3.8 (3.3)
  Endpoint visit; n=27, 22, 18 | 3.9 (3.2) | 3.5 (2.6) | 4.0 (2.8)

56. Other Pre Specified Outcome: UPDRS Part II Score, up to Month 36
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. For Parts I-III and Total Score, each question is measured on a 5-point scale of 0 (normal or no disease effect) to 4 (maximum negative effect). Part II score is the sum of answers to 'Activities of Daily Living' questions, with a score range from 0-52. Higher scores are associated with more disability.
Time Frame: Months 0, 3, 6, 9, 18, 24, 30, 36, endpoint (last non-missing value assigned to treatment for the participant)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Month 0; n=27, 22, 18 | 12.3 (5.1) | 13.7 (6.3) | 15.4 (5.9)
  Month 3; n=24, 22, 18 | 12.0 (5.7) | 12.8 (7.1) | 15.0 (5.8)
  Month 6; n=25, 22, 18 | 12.4 (6.7) | 13.4 (6.7) | 14.3 (4.4)
  Month 9; n=25, 20, 17 | 11.8 (6.9) | 13.0 (5.5) | 14.4 (5.2)
  Month 18; n=24, 20, 17 | 13.3 (7.2) | 12.9 (6.6) | 15.6 (5.8)
  Month 24; n=23, 18, 15 | 12.9 (7.7) | 12.2 (6.2) | 17.2 (5.3)
  Month 30; n=23, 17, 13 | 14.0 (8.5) | 14.6 (7.3) | 16.9 (6.3)
  Month 36; n=21, 16, 12 | 13.9 (8.4) | 14.6 (5.4) | 16.8 (8.2)
  Endpoint visit; n=27, 22, 18 | 14.6 (7.9) | 15.7 (6.4) | 17.3 (7.0)

57. Other Pre Specified Outcome: UPDRS Part III Score, up to Month 36
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. For Parts I-III and Total Score, each question is measured on a 5-point scale of 0 (normal or no disease effect) to 4 (maximum negative effect). Part III score is the sum of answers to 'Motor Examination' questions, with a score range from 0-108. Higher scores are associated with more disability.
Time Frame: Months 0, 3, 6, 9, 18, 24, 30, 36, endpoint (last non-missing value assigned to treatment for the participant)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Month 0; n=27, 22, 18 | 22.0 (9.7) | 23.4 (11.1) | 22.4 (9.8)
  Month 3; n=24, 22, 18 | 21.6 (11.5) | 22.9 (11.3) | 21.9 (9.5)
  Month 6; n=25, 20, 18 | 21.5 (14.1) | 22.8 (9.9) | 22.6 (8.6)
  Month 9; n=25, 20, 17 | 19.9 (12.4) | 21.9 (8.1) | 22.9 (11.8)
  Month 18; n=24, 20, 16 | 21.3 (12.6) | 21.7 (9.3) | 23.3 (11.1)
  Month 24; n=23, 18, 15 | 21.4 (14.2) | 18.2 (9.8) | 25.4 (9.2)
  Month 30; n=23, 17, 13 | 23.1 (15.6) | 22.6 (11.5) | 24.0 (12.1)
  Month 36; n=21, 16, 12 | 22.0 (17.2) | 22.2 (7.9) | 28.0 (15.8)
  Endpoint visit; n=27, 22, 17 | 23.1 (15.8) | 24.1 (9.8) | 28.6 (13.6)

58. Other Pre Specified Outcome: UPDRS Part IV Score, up to Month 36
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. For Part IV, questions are measured on a 5-point scale of 0 (normal or no disease effect) to 4 (maximum negative effect) or 2-point scale (0 or 1). Part IV score is the sum of answers to 'Complications of Therapy' questions, with a score range from 0-23. Higher scores are associated with more disability.
Time Frame: Months 0, 3, 6, 9, 18, 24, 30, 36, endpoint (last non-missing value assigned to treatment for the participant)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Month 0; n=27, 22, 18 | 6.5 (2.7) | 7.1 (3.4) | 7.2 (3.0)
  Month 3; n=24, 22, 18 | 6.3 (2.9) | 7.8 (3.1) | 6.7 (3.4)
  Month 6; n=25, 22, 18 | 6.5 (2.7) | 7.1 (2.8) | 7.7 (3.2)
  Month 9; n=25, 20, 17 | 6.1 (3.3) | 7.3 (3.3) | 7.5 (4.2)
  Month 18; n=24, 20, 17 | 6.5 (3.3) | 7.0 (3.2) | 7.6 (2.8)
  Month 24; n=23, 18, 15 | 6.3 (4.3) | 6.8 (3.6) | 6.6 (2.5)
  Month 30; n=22, 17, 13 | 6.2 (3.7) | 6.6 (3.3) | 6.5 (2.8)
  Month 36; n=21, 16, 12 | 6.4 (3.0) | 6.4 (2.4) | 5.5 (1.8)
  Endpoint visit; n=26, 22, 18 | 6.5 (3.0) | 7.5 (3.0) | 6.7 (2.7)

59. Other Pre Specified Outcome: EQ-5D Descriptive Systems Summary Index Score, up to Month 36
Description: The EQ-5D is a participant-answered questionnaire scoring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that essentially attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.11 to 1.00 with positive change indicating improvement.
Time Frame: Months 0, 3, 6, 9, 18, 24, 30, 36, endpoint (last non-missing value assigned to treatment for the participant)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Month 0; n=27, 22, 18 | 0.67 (0.27) | 0.68 (0.27) | 0.62 (0.24)
  Month 3; n=24, 22, 18 | 0.61 (0.30) | 0.70 (0.29) | 0.57 (0.32)
  Month 6; n=25, 21, 18 | 0.64 (0.26) | 0.71 (0.22) | 0.57 (0.32)
  Month 9; n=25, 20, 17 | 0.61 (0.33) | 0.66 (0.23) | 0.59 (0.30)
  Month 18; n=24, 20, 16 | 0.64 (0.23) | 0.66 (0.34) | 0.53 (0.35)
  Month 24; n=21, 18, 15 | 0.58 (0.33) | 0.67 (0.26) | 0.47 (0.32)
  Month 30; n=22, 17, 12 | 0.55 (0.28) | 0.69 (0.19) | 0.52 (0.28)
  Month 36; n=21, 15, 11 | 0.52 (0.31) | 0.57 (0.28) | 0.51 (0.25)
  Endpoint visit; n=26, 22, 17 | 0.54 (0.31) | 0.60 (0.25) | 0.46 (0.33)

60. Other Pre Specified Outcome: EQ-5D Visual Analog Scale (VAS) Score, up to Month 36
Description: The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where 100 is the 'best imaginable health state' and 0 is the 'worst imaginable health state.'
Time Frame: Months 0, 3, 6, 9, 18, 24, 30, 36, endpoint (last non-missing value assigned to treatment for the participant)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Number analyzed (Participants) | 27 | 22 | 18
units on a scale
  Month 0; n=27, 22, 18 | 0.68 (0.18) | 0.65 (0.18) | 0.58 (0.23)
  Month 3; n=24, 22, 18 | 0.65 (0.19) | 0.63 (0.18) | 0.58 (0.20)
  Month 6; n=25, 21, 18 | 0.60 (0.22) | 0.65 (0.16) | 0.59 (0.18)
  Month 9; n=25, 20, 17 | 0.68 (0.14) | 0.69 (0.15) | 0.58 (0.19)
  Month 18; n=24, 20, 16 | 0.62 (0.20) | 0.60 (0.20) | 0.55 (0.27)
  Month 24; n=21, 17, 15 | 0.64 (0.18) | 0.60 (0.20) | 0.63 (0.12)
  Month 30; n=22, 17, 12 | 0.56 (0.20) | 0.67 (0.14) | 0.65 (0.17)
  Month 36; n=21, 15, 11 | 0.56 (0.17) | 0.61 (0.18) | 0.62 (0.19)
  Endpoint visit; n=26, 22, 17 | 0.57 (0.16) | 0.61 (0.17) | 0.57 (0.21)

ADVERSE EVENTS:
Time Frame: Events presented are treatment-emergent (those with a start date beyond or equal to first day of study treatment but within 7 days [for adverse events] or 30 days [for serious adverse events] after last study drug intake). Treatment period was 36 months.
Arm/Group | Duodopa Naïve | Duodopa Non-naïve < 2 Years | Duodopa Non-naïve ≥ 2 Years
Serious Adverse Events (participants affected / at risk) | 24/36 | 17/22 | 14/18
Other Adverse Events (participants affected / at risk) | 29/36 | 22/22 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duodopa Naïve (N=36) | Duodopa Non-naïve < 2 Years (N=22) | Duodopa Non-naïve ≥ 2 Years (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 1
Gait disturbance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0
Therapeutic response decreased (General disorders) | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 3 | 1 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gastric ulcer helicobacter (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device breakage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Device connection issue (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 3 | 1 | 1
Device occlusion (Injury, poisoning and procedural complications) | 2 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 2
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0 | 2
Medical device pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0
Electrocardiogram rr interval prolonged (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 2 | 1 | 2
Dystonia (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Hyperkinesia (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
On and off phenomenon (Nervous system disorders) | 1 | 1 | 0
Parkinson's disease (Nervous system disorders) | 2 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 4 | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep brain stimulation (Surgical and medical procedures) | 0 | 1 | 0
Device therapy (Surgical and medical procedures) | 0 | 0 | 1
Drug therapy changed (Surgical and medical procedures) | 0 | 1 | 1
Medical device change (Surgical and medical procedures) | 9 | 9 | 3
Medical device implantation (Surgical and medical procedures) | 0 | 1 | 0
Medical device removal (Surgical and medical procedures) | 0 | 3 | 0
Pelvic floor repair (Surgical and medical procedures) | 1 | 0 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 0 | 1
Therapy regimen changed (Surgical and medical procedures) | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duodopa Naïve (N=36) | Duodopa Non-naïve < 2 Years (N=22) | Duodopa Non-naïve ≥ 2 Years (N=18)
Anaemia (Blood and lymphatic system disorders) | 6 | 4 | 2
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 8 | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Implant site inflammation (General disorders) | 0 | 1 | 0
Implant site pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 2
Candidiasis (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 4 | 6 | 4
Erysipelas (Infections and infestations) | 0 | 0 | 1
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 4 | 4
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device connection issue (Injury, poisoning and procedural complications) | 2 | 0 | 0
Device dislocation (Injury, poisoning and procedural complications) | 7 | 8 | 5
Device occlusion (Injury, poisoning and procedural complications) | 3 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 2
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Medical device pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 2 | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood amino acid level increased (Investigations) | 0 | 0 | 1
Blood folate decreased (Investigations) | 1 | 0 | 1
Blood homocysteine increased (Investigations) | 2 | 4 | 6
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0
Cerebrospinal fluid white blood cell count decreased (Investigations) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 3 | 0 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 0 | 1
Residual urine volume (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 2 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 4 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypovitaminosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1 | 1
Dementia (Nervous system disorders) | 3 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Dystonia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 7 | 4 | 2
Hallucination (Psychiatric disorders) | 7 | 2 | 2
Insomnia (Psychiatric disorders) | 6 | 3 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 6 | 2
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 3 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2 | 1
Prostatism (Reproductive system and breast disorders) | 0 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 6 | 7 | 2
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cardiac operation (Surgical and medical procedures) | 1 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0
Eye operation (Surgical and medical procedures) | 0 | 1 | 0
Knee operation (Surgical and medical procedures) | 0 | 1 | 0
Medical device change (Surgical and medical procedures) | 6 | 5 | 1
Medical device removal (Surgical and medical procedures) | 1 | 0 | 0
Prostatic operation (Surgical and medical procedures) | 0 | 0 | 1
Shoulder operation (Surgical and medical procedures) | 1 | 0 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0 | 0
Tendon operation (Surgical and medical procedures) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.